

## PROTOCOL: SHP465-308

TITLE: A Phase 3, Open-label, Multicenter, 12-Month Safety and Tolerability

Study of SHP465 in Children Aged 4 to 12 Years Diagnosed with

Attention-deficit/Hyperactivity Disorder

**DRUG:** SHP465, mixed salts of a single-entity amphetamine

66,329 IND:

**EUDRACT NO.:** Non-EUDRACT

**SPONSOR:** Shire Development LLC

300 Shire Way, Lexington, MA 02421 USA

PRINCIPAL/ COORDINATING MD

**INVESTIGATOR:** 

**PROTOCOL HISTORY:** 

Version 2.0: 18 May 2018

This document contains confidential and proprietary information of Shire and is disclosed pursuant to confidentiality and non-disclosure obligations. This information should be used solely for the purposes for which it was provided and should not be copied, shared with, or disclosed to any third party without the express written consent of Shire.

# PROTOCOL SIGNATURE PAGE

| Signature: | Date: |
|---|---|
| The second secon | |
| Investigator's Acknowledgement | t |
| I have read this protocol for Shire S | Study SHP465-308. |
| | ticenter, 12-Month Safety and Tolerability Study of SHP46 nosed with Attention-deficit/Hyperactivity Disorder |
| I have fully discussed the objective sponsor's representative. | es of this study and the contents of this protocol with the |
| other than to those directly involve without written authorization from | n this protocol is confidential and should not be disclosed, ed in the execution or the scientific/ethical review of the state the sponsor. It is, however, permissible to provide the subject in order to obtain their consent to participate. |
| subject to ethical and safety consid | ding to this protocol and to comply with its requirements, lerations and guidelines, and to conduct the study in neil for Harmonisation guidelines on Good Clinical Practic requirements. |
| I understand that failure to comply<br>termination of my participation as | with the requirements of the protocol may lead to the an investigator for this study. |
| time for whatever reason; such a de | decide to suspend or prematurely terminate the study at any ecision will be communicated to me in writing. Conversely execution of the study I will communicate my intention sor. |
| Investigator Name and Address: | |
| (please hand print or type) | |
| - | |

# **EMERGENCY CONTACT INFORMATION**

In the event of an SAE, the investigator must fax or e-mail the Shire Clinical Trial Serious Adverse Event Form within 24 hours to the Shire Global Drug Safety Department. Applicable fax numbers and e-mail address can be found on the form (sent under separate cover). A copy of the Shire Clinical Trial Serious Adverse Event Form must also be sent to the CRO/Shire medical monitor by e-mail using the details below.

| the Shire Clinical Trial S<br>monitor by e-mail using | derious Adverse Event Form must also be sent to the CRO/Shire med the details below. |
|---|---|
| E-mail address: | (electronic query submission site) |
| | related issues during normal business hours 8AM-5PM eastern stigator must contact the PPD medical monitor: |
| , MD | |
| Phone: | |
| Mobile: | (callers will be transferred to the medical monitor's cell phone) |
| For protocol- or safety-recontact the PPD medical | elated issues <u>outside of normal business hours</u> , the investigator must monitor: |
| Phone: | |

# PRODUCT QUALITY COMPLAINTS

Investigators are required to report investigational product quality complaints to Shire within 24 hours. This includes any instances wherein the quality or performance of a Shire product (marketed or investigational) does not meet expectations (eg, inadequate or faulty closure, product contamination) or that the product did not meet the specifications defined in the application for the product (eg, wrong product such that the label and contents are different products). For instructions on reporting AEs related to product complaints, see Section 8.

Please use the information as follows as applicable to report the Product Quality Complaint:

| Origin of Product Quality Complaint | Email Address |
|-------------------------------------|---------------|
| North and South America | |

Telephone numbers (provided for reference if needed):

Shire, Lexington, MA (USA)

# AMENDMENT SUMMARY AND RATIONALE

Noteworthy changes to the protocol are captured in the table below. Additional minor revisions in grammar, spelling, punctuation, and format were made for clarity and are not reflected in the summary of changes.

## **Summary of Changes from Previous Version**

| Protocol Amendments | | |
|---|---|---|
| Summary of Change(s) Since Last Version of Approved Protocol | | |
| Amendment Number | Amendment Date | Global/Country/Site Specific |
| 4 | 18 May 2018 | Global |
| Description | n of Change | Section(s) Affected by Change |
| | en increased to approximately 145 in | Study Synopsis |
| subjects from SHP465-112. | arollment status and future rollover of | Section 3.1 |
| | | Section 9.6 |
| Administrative changes were incorp | orated per Administrative Change | Schedule of Assessments |
| Memo 1, dated 17 Oct 2017: | | Section 4.2.2 |
| Physical exam and AE coll- of Assessments for Group I | ection timing corrected in Schedule | Section 7.2.3.2 |
| | | Section 7.2.3.6 |
| <ul> <li>Clarification of timing of urine drug screen and clarification of<br/>maximum storage time for blood and urine samples</li> </ul> | | Section 8.1.6 |
| <ul> <li>Clarification of need to report pregnancies in the partners of male subjects</li> <li>Clarification of male contraception requirements</li> </ul> | | |
| Administrative changes were incorporated per Administrative Change | | Protocol title page |
| Memo 2, dated 27 Nov 2017: | SELECTION SHEETING BY HE CASE OF THE SHEETING | Section 3.1 |
| | and Flow Chart" for Groups A and B en placed under the correct titles. | |
| The name of the Principal/0 MD, is now supple | | |
| Administrative changes were incorporated per Administrative Change Memo 3, dated 22 Mar 2018: | | Section 7.2.3.6 |
| The following lab evaluations were clarified: "T4," to "Thyroxine, Free"; "Uric acid" to "Urate"; "Bands," to "Neutrophils Band Forms"; "Nitrate," to "Nitrite" | | |

# TABLE OF CONTENTS

| PF | ROTOCOL S | IGNATURE PAGE | 2 |
|---|---|---|---|
| EN | MERGENCY | CONTACT INFORMATION | 3 |
| PF | RODUCT QU | ALITY COMPLAINTS | 4 |
| Al | MENDMENT | SUMMARY AND RATIONALE | 5 |
| TA | ABLE OF CO | NTENTS | 6 |
| LI | ST OF TABI | LES | 10 |
| LI | ST OF FIGU | RES | 10 |
| Al | BBREVIATION | ONS | 11 |
| SI | TUDY SYNO | PSIS | 12 |
| SI | TUDY SCHE | DULES | 17 |
| 1 | BACKGRO | OUND INFORMATION | 23 |
| | 1.1 In | dication and Current Treatment Options | 23 |
| | 1.2 Pr | oduct Background and Clinical Information | 24 |
| 2 | STUDY O | BJECTIVES AND PURPOSE | 25 |
| | 2.1 Ra | ationale for the Study | 25 |
| | 2.2 St | udy Objectives | 25 |
| | 2.2.1 I | Primary Objective | 25 |
| | 2.2.2 | Secondary Objectives | 25 |
| 3 | | ESIGN | |
| | | udy Design and Flow Chart | |
| | | uration and Study Completion Definition | |
| | | tes and Regions | |
| 4 | | OPULATION | |
| | | clusion Criteria | |
| | | xclusion Criteria | |
| | | Female Contraception | |
| | | Male Contraception | |
| | | iscontinuation of Subjects | |
| | | Management of Blood Pressure and Pulse During the Study | |
| | 4.3.1 | | |
| | 4.3.1 | | |
| | | Reasons for Discontinuation | |
| _ | | Subjects "Lost to Follow-up" Prior to Last Scheduled Visit | |
| 5 | | ID CONCOMITANT TREATMENT | |
| | | ior Treatment | |
| | 5.2 Co | oncomitant Treatment | 34 |

| Study Protocol | Amendment 2 |
|----------------|-------------|
| SHP465-308 | |

| 10 | 3.6 | 2010 |
|----|-----|------|
| 18 | May | 2018 |

| | | | -, |
|---|---|---|---|
| | 5.2.1 | Permitted Treatment. | 34 |
| | 5.2.2 | Prohibited Treatment | 34 |
| 6 | INVEST | IGATIONAL PRODUCT | 36 |
| | 6.1 | Identity of Investigational Product | 36 |
| | 6.1.1 | Blinding the Treatment Assignment | 36 |
| | 6.2 | Administration of Investigational Product(s) | 36 |
| | 6.2.1 | Interactive Response Technology for Investigational Product Management | 36 |
| | 6.2.2 | Allocation of Subjects to Treatment | 36 |
| | 6.2.3 | Dosing | 36 |
| | 6.2.4 | Unblinding the Treatment Assignment | 37 |
| | 6.3 | Labeling, Packaging, Storage, and Handling | 37 |
| | 6.3.1 | Labeling | 37 |
| | 6.3.2 | Packaging | 38 |
| | 6.3.3 | Storage | 38 |
| | 6.4 | Drug Accountability | 39 |
| | 6.5 | Subject Compliance | 40 |
| 7 | STUDY | PROCEDURES | 41 |
| | 7.1 | Study Schedule | 41 |
| | 7.1.1 | Screening and Washout Period (Group A and Group B) | 41 |
| | 7. | 1.1.1 Screening Visit (Visit 1) for Group B | 42 |
| | 7. | 1.1.2 Washout Telephone Call (Group B) | 43 |
| | 7. | 1.1.3 Baseline Visit (Visit 2) Group A | |
| | 7. | 1.1.4 Baseline Visit (Visit 2) Group B | 44 |
| | 7.1.2 | Treatment Period (Group A and Group B) | 45 |
| | 7. | 1.2.1 Treatment Period (Visits 5 to 16/Early Termination) | |
| | 7.1.3 | Safety Follow-up Period (Group A and Group B) | 46 |
| | 7.1.4 | Additional Care of Subjects After the Study | 47 |
| | 7.2 | Study Evaluations and Procedures | |
| | 7.2.1 | Demographic and Other Baseline Characteristics | 47 |
| | 7. | 2.1.1 Mini International Neuropsychiatric Interview for Children and Adolescents | 47 |
| | 7.2.2 | Efficacy | |
| | | 2.2.1 The ADHD-Rating Scale-5 | |
| | | 2.2.2 Clinical Global Impression | |
| | 7.2.3 | • | |
| | | 2.3.1 Medical and Medication History | |
| | | 2.3.2 Physical Examination (Including Height and Weight) | |
| | | 2.3.3 Adverse Event Collection | |
| | /. | | 50 |

| Study Protocol | Amendment 2 |
|----------------|-------------|
| SHP465-308 | |

| 18 May 2 | 018 |
|----------|-----|
|----------|-----|

| | 7. | 2.3.4 Vital Signs | 50 |
|---|---|---|---|
| | 7. | 2.3.5 Height and Weight | |
| | 7. | 2.3.6 Clinical Laboratory Evaluations | 51 |
| | 7. | 2.3.7 Pregnancy Test | 53 |
| | 7. | 2.3.8 Electrocardiogram | 55 |
| | 7. | 2.3.9 Post Sleep Questionnaire | 55 |
| | 7. | 2.3.10 Children's Sleep Habits Questionnaire | 55 |
| | 7. | 2.3.11 Columbia-Suicide Severity Rating Scale-Baseline Version | 56 |
| | 7. | 2.3.12 Suitability of the Subject to Remain in the Study | 56 |
| | 7.2.4 | Volume of Blood to Be Drawn From Each Subject | 57 |
| 8 | ADVER | SE AND SERIOUS ADVERSE EVENTS ASSESSMENT | 58 |
| | 8.1 | Definition of Adverse Events, Period of Observation, Recording of Adverse Events | 58 |
| | 8.1.1 | Severity Categorization | |
| | 8.1.2 | Relationship Categorization | |
| | 8.1.3 | Outcome Categorization | |
| | 8.1.4 | Symptoms of the Disease Under Study | 59 |
| | 8.1.5 | Clinical Laboratory and Other Safety Evaluations | 59 |
| | 8.1.6 | Pregnancy | 60 |
| | 8.1.7 | Abuse, Misuse, Overdose, and Medication Error | 60 |
| | 8.2 | Serious Adverse Event Procedures | 61 |
| | 8.2.1 | Reference Safety Information | 61 |
| | 8.2.2 | Reporting Procedures | 61 |
| | 8.2.3 | Serious Adverse Event Definition | 62 |
| | 8.2.4 | Serious Adverse Event Collection Time Frame | 62 |
| | 8.2.5 | Serious Adverse Event Onset and Resolution Dates | 63 |
| | 8.2.6 | Fatal Outcome | 63 |
| | 8.2.7 | Regulatory Agency, Institutional Review Board, Ethics Committee, and Site Reporting | 63 |
| 9 | DATA N | MANAGEMENT AND STATISTICAL METHODS | 64 |
| | 9.1 | Data Collection | 64 |
| | 9.2 | Clinical Data Management | 64 |
| | 9.3 | Data Handling Considerations | 64 |
| | 9.4 | Statistical Analysis Process | 64 |
| | 9.5 | Planned Interim Analysis, Adaptive Design, and Data Monitoring Committee | 65 |
| | 9.5.1 | Interim Analysis | 65 |
| | 9.5.2 | Data Monitoring Committee | |
| | 9.6 | Sample Size Calculation and Power Considerations | 65 |

| Stu | re<br>dy Protoco | ol Amendment 2 | Page 9 |
|---|---|---|---|
| | P465-308 | of Amendment 2 | 18 May 2018 |
| | 9.7 | Study Population | 65 |
| | 9.8 | Efficacy Analyses | 65 |
| | 9.9 | Safety Analyses | 66 |
| 10 | SPONS | OR'S AND INVESTIGATOR'S RESPONSIBILITIES | 68 |
| | 10.1 | Sponsor's Responsibilities | 68 |
| | 10.1. | .1 Good Clinical Practice Compliance | 68 |
| | 10.1. | .2 Public Posting of Study Information | 68 |
| | 10.1. | .3 Submission of Summary of Clinical Study Report to Competent Autloof Member States Concerned and Ethics Committees | |
| | 10.1. | .4 Study Suspension, Termination, and Completion | |
| | 10.2 | Investigator's Responsibilities | |
| | 10.2. | .1 Good Clinical Practice Compliance | |
| | | .2 Protocol Adherence and Investigator Agreement | |
| | | .3 Documentation and Retention of Records | |
| | 1 | 10.2.3.1 Case Report Forms | 70 |
| | 1 | 10.2.3.2 Recording, Access, and Retention of Source Data and Stud Documents | • |
| | 1 | 10.2.3.3 Audit/Inspection | 70 |
| | 1 | 10.2.3.4 Financial Disclosure | 71 |
| | 10.2. | .4 Compliance to all Local, State, and National Controlled-substance | |
| | | Biohazard and Infectious Disease Regulations and Legislation | |
| | 10.3 | Ethical Considerations | |
| | | .1 Informed Consent | |
| | | .2 Institutional Review Board or Ethics Committee | |
| | 10.4 | Privacy and Confidentiality | |
| | 10.5 | Study Results/Publication Policy | |
| 11 | | ENCES | |
| 12 | | IDICES | |
| | PENDIX | | |
| Aŀ | PENDIX | | |
| | Appendi | | |
| | Appendi | | |
| | Appendi | | |
| | Appendi | | |
| A T | Appendi | | |
| Al | PENDIX | SCALES AND ASSESSMENTS | 88 |

# LIST OF TABLES

| Table 1: | Schedule of Assessments for Group A | 17 |
|---|---|---|
| Table 2: | Schedule of Assessments for Group B | 20 |
| Table 3: | Common Excluded Treatments and Associated Washout<br>Period - Relative to Baseline Visit (Visit 2) | 35 |
| Table 4: | Volume of Blood to Be Drawn From Each Subject | 57 |
| | LIST OF FIGURES | |
| Figure 1: | Study Design Flow Chart for Group A | 26 |
| Figure 2: | Study Design Flow Chart for Group B | 27 |

Study Protocol Amendment 2 SHP465-308

18 May 2018

## **ABBREVIATIONS**

ADHD attention-deficit/hyperactivity disorder

ADHD-RS-5 Attention-deficit/Hyperactivity Disorder Rating Scale 5

AE adverse event BMI body mass index

CGI Clinical Global Impressions

CGI-I Clinical Global Impressions – Improvement
CGI-S Clinical Global Impressions – Severity of Illness

CRF case report form

CRO contract research organization

CSHQ Children's Sleep Habits Questionnaire
C-SSRS Columbia-Suicide Severity Rating Scale

DMC data monitoring committee

DSM-5 Diagnostic and Statistical Manual of Mental Disorders, 5th edition

EC Ethics Committee
ECG electrocardiogram
ET early termination
FAS full analysis set

FDA Food and Drug Administration

GCP Good Clinical Practice

HIPAA Health Insurance Portability and Accountability Act

ICH International Council for Harmonisation

IRB Institutional Review Board

IWRS interactive web response system LAR legally authorized representative

MINI-KID Mini International Neuropsychiatric Interview for Children and

Adolescents

PSQ Post Sleep Questionnaire

PK pharmacokinetic(s)
SAE serious adverse event
SAP statistical analysis plan

TEAE treatment-emergent adverse event

US United States

## STUDY SYNOPSIS

**Protocol number:** SHP465-308 **Drug:** SHP465, mixed salts of a single-entity amphetamine

**Title of the study:** A Phase 3, Open-label, Multicenter, 12-Month, Safety and Tolerability Study of SHP465 in Children Aged 4 to 12 Years Diagnosed with Attention-deficit/Hyperactivity Disorder

#### Number of subjects (total and for each treatment arm):

Approximately 145 subjects will be enrolled into this study to ensure 60 subjects complete at least 6 months of study treatment. Subjects will enroll into this study either directly or from antecedent studies SHP465-112 or SHP465-309. The sample size was established to provide long term safety data in this population and will include at least 40 subjects aged 4-5 years at the time of informed consent in the antecedent trial or this trial, if directly enrolled.

**Investigators:** Multicenter study

**Sites and region:** Approximately 50 sites in the United States (US)

Study period (planned): 2017-2019 | Clinical phase: 3

#### **Objectives:**

**Primary:** To evaluate the long-term safety and tolerability of SHP465 at 6.25 mg administered as a daily morning dose in children aged 4-12 years, inclusive, diagnosed with Attention-deficit/Hyperactivity Disorder (ADHD).

The evaluation of safety and tolerability will be based on the occurrence of treatment-emergent adverse events (TEAEs), evaluation of vital signs (systolic and diastolic blood pressure and pulse), weight, height, body mass index (BMI); clinical laboratory and electrocardiogram (ECG) results; sleep assessment (Post Sleep Questionnaire [PSQ] and Children's Sleep Habits Questionnaire [CSHQ]); and responses to the Columbia-Suicide Severity Rating Scale (C-SSRS).

#### Secondary:

- 1. To describe the long-term efficacy of SHP465 using the clinician-administered ADHD Rating Scale 5 (ADHD-RS-5) Child, Home Version.
- 2. To describe the long-term efficacy of SHP465 using the Clinical Global Impressions–Improvement (CGI-I) scale.

#### **Rationale:**

The purpose of the study is to evaluate the long-term safety of SHP465 in children aged 4 to 12 years diagnosed with ADHD. Results from this study will provide important information on the long-term safety, tolerability, and efficacy of SHP465 at lower doses in the preschool/pediatric ADHD population.

#### Investigational product, dose, and mode of administration:

SHP465 will be provided as 6.25 mg capsules.

The parent/legally authorized representative (LAR) will be instructed to dispense 1 capsule to the subject daily throughout the study at 7:00 AM ( $\pm 2$  hours). SHP465 will be administered in 1 of the following ways:

- Swallow SHP465 capsules whole, or
- Open capsule and sprinkle the entire contents on applesauce.

The sprinkled applesauce should be consumed immediately; it should not be stored. Subjects should take the sprinkled applesauce in its entirety without chewing.

#### Methodology:

This study is a Phase 3 long-term, open-label, multicenter, safety and tolerability study in children (aged 4-12 years, inclusive, at the time of consent was obtained in the antecedent study [SHP465-112 or SHP465-309] or at the time of consent into this study if directly enrolled) with ADHD.

Subjects enrolled in this study will be divided into 2 groups based on participation in antecedent studies as follows:

- Subjects in Group A are those who have been rolled-over from antecedent studies (SHP465-112 or SHP465-309). These subjects do not need additional screening and washout procedures.
- Subjects in Group B will be newly enrolled subjects who will be required to undergo full screening and
  washout before enrollment.

Subjects in Group A will participate in the following 2 study periods: (1) treatment period and (2) safety follow-up. Subjects in Group B will participate in the following 3 study periods: (1) screening and washout, (2) treatment period, and (3) safety follow-up.

For subjects in Group A, the last visit of the antecedent study, SHP465-112 or SHP465-309, will serve as the baseline visit (Visit 2) for this study. For subjects in Group B, a screening visit will precede a washout period.

Subjects aged 4-12 years will receive SHP465 at a fixed dose of 6.25 mg.

Subjects in both groups will be treated and evaluated for 12 months, and visit the site up to 15 times for subjects in Group A and up to 16 times for subjects in Group B.

The investigator or designee must obtain written informed consent from the subject's parent/LAR and documentation of assent (if applicable) by the subject before any protocol-related procedure is performed. Procedures performed at each visit for all subjects are defined in the Study Schedules: Table 1 (Group A) and Table 2 (Group B).

#### Inclusion and exclusion criteria:

#### **Inclusion Criteria:**

The subject will not be considered eligible for the study without meeting all of the following criteria (including test results):

- 1. Subject is male or female aged 4 to 12 years, inclusive, at the time of consent for antecedent SHP465 trials (SHP465 112 or SHP465-309) in the ADHD population or at the time of consent for directly enrolled subjects into this study.
- 2. Subject's parent or legally authorized representative (LAR) must provide signature of informed consent, and there must be documentation of assent (if applicable) by the subject in accordance with the International Council on Harmonization (ICH) Good Clinical Practice (GCP) Guideline E6 (1996) and any updates and applicable regulations, before completing any study-related procedures.
- 3. Subject and parent/LAR are willing and able to comply with all of the testing and requirements defined in the protocol, including oversight of morning dosing. Specifically, the same parent/LAR should be available daily to dispense the dose of investigational product for the duration of the study.
- 4. For subjects in Group A:
  - Subject enrolled in the antecedent study SHP465-112 must have completed treatment period and the pharmacokinetic (PK) sample collection (at the dose of 6.25 mg) without incidence of a clinically significant TEAE.
  - Subject enrolled in the antecedent study SHP465-309 must have completed the treatment period without reporting a clinically significant TEAE that would preclude subsequent exposure to SHP465.
- 5. For subjects in Group B (directly enrolled subjects), the following criteria must be met:
  - Subject meets the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for a primary diagnosis of ADHD (any subtype) based on a detailed psychiatric evaluation using the Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-KID)

- Subject aged 4 to 5 years has an ADHD-RS-5 Child Version Total score of ≥28 (boys) or ≥24 (girls) at baseline (Visit 2)
- Subject aged 6 to 12 years has an ADHD-RS-5 Child, Home Version Total score of ≥28 at baseline (Visit 2)
- Subject has a Clinical Global Impression—Severity of Illness score (CGI-S) ≥4 at baseline (Visit 2)
- Subject has previously undergone an adequate course of nonpharmacological treatment based on
  investigator judgment (aged 4-5 year olds) OR the subject is not completely satisfied with current
  adequate course of ADHD therapy (aged 6-12 year olds), OR the subject has a severe enough
  condition to consider enrollment without undergoing prior nonpharmacological treatment, based on
  investigator judgment.
- Subject functions as an age-appropriate level intellectually, based on investigator judgment.
- 6. Subject who is a female and of child-bearing potential must not have a positive serum beta human chorionic gonadotropin pregnancy test at the screening visit (Visit 1) and must have a negative urine pregnancy test at the baseline visit (Visit 2) and agree to comply with any applicable contraceptive requirements of the protocol.
- 7. Subject has lived with the same parent/LAR for at least 6 months.

#### **Exclusion Criteria:**

Subjects will be excluded from the study if any of the following exclusion criteria are met at baseline (Visit 2) for Group A or at screening (Visit 1) and/or baseline (Visit 2) for Group B. These criteria apply to all subjects regardless of participation in an antecedent trial:

- 1. Subject was terminated from an antecedent SHP465 trial for noncompliance and/or had a serious TEAE during any previous SHP465 trial.
- 2. Subject is required to or is anticipated to take any medication that has central nervous system effects or affects performance, such as sedating antihistamines and decongestant sympathomimetics, or is a monoamine oxidase inhibitor. Stable use of bronchodilator inhalers is not exclusionary.
- 3. Subject has a concurrent chronic or acute illness (such as severe allergic rhinitis or an infectious process requiring antibiotics), disability, or other condition that might confound the results of safety assessments conducted in the study or that might increase risk to the subject. Similarly, the subject will be excluded if he or she has any additional condition(s) that, in the investigator's opinion, would prohibit the subject from completing the study or would not be in the best interest of the subject. The additional condition(s) would include any significant illness or unstable medical condition that could lead to difficulty complying with the protocol. Mild, stable asthma is not exclusionary.
- 4. Subject has a documented allergy, hypersensitivity, or intolerance to amphetamine or to any excipients in the investigational product.
- 5. Subject has a known family history of sudden cardiac death or ventricular arrhythmia.
- 6. Subject has a blood pressure measurement ≥95<sup>th</sup> percentile for age, sex, and height at screening (Visit 1) and/or baseline (Visit 2).
- 7. Subject has a height ≤5th percentile for age and sex at screening (Visit 1) and/or baseline (Visit 2).
- 8. Subject has a weight ≤5th percentile for age and sex at screening (Visit 1) and/or baseline (Visit 2).
- 9. Subject has a known history of symptomatic cardiovascular disease, structural cardiac abnormality, cardiomyopathy, serious heart rhythm abnormalities, or other serious cardiac conditions placing them at increased vulnerability to the sympathomimetic effects of a stimulant drug.
- 10. Subject has a history of seizures (other than infantile febrile seizures).
- 11. Subject has failed to fully respond, based on investigator judgment, to an adequate course of amphetamine therapy.
- 12. Subject is taking any medication that is excluded per the protocol.

- 13. Subject had any clinically significant ECG or clinical laboratory abnormalities at the screening (Visit 1) and/or baseline visit (Visit 2).
- 14. Subject has current abnormal thyroid function, defined as abnormal thyroid-stimulating hormone and thyroxine at the screening (Visit 1) and/or baseline visit (Visit 2). Treatment with a stable dose of thyroid medication for at least 3 months is permitted.
- 15. Subject has a current, controlled (requiring medication or therapy) or uncontrolled, comorbid psychiatric disorder including, but not limited to, any of the following comorbid Axis I disorders and Axis II disorders:
  - Post-traumatic stress disorder or adjustment disorder
  - Bipolar disorder, psychosis, schizophrenia or family history of these disorders
  - Pervasive developmental disorder
  - Obsessive-compulsive disorder
  - Serious tic disorder, or a family history of Tourette disorder
  - Any other disorder that in the opinion of the investigator contraindicates SHP465 or amphetamine treatment or confounds efficacy or safety assessments
- 16. Subject has a primary sleep disorder (eg, sleep apnea, narcolepsy)
- 17. Subject has a history or is currently diagnosed with an eating disorder
- 18. Subject is currently considered a suicide risk in the opinion of the investigator, has previously made a suicide attempt, or has a prior history of or currently demonstrating suicidal ideation.
- 19. Subject has a history of physical, sexual, or emotional abuse.
- 20. Subject has initiated behavioral therapy within 1 month before baseline (Visit 2). Subject may not initiate behavioral therapy during the study.
- 21. Subject has a clinically important abnormality on the urine drug and alcohol screen (except for the subject's current ADHD stimulant, if applicable) at screening (Visit 1) or baseline (Visit 2).
- 22. Subject is female and pregnant or lactating.
- 23. Subject cannot swallow a pill and/or applesauce or has an allergy to applesauce.

#### Maximum duration of subject involvement in the study:

Planned duration of screening/washout:

- For Group A (subjects from antecedent studies): None
- For Group B (directly enrolled subjects): up to 32 days

Planned duration of treatment:

- For Group A (subjects from antecedent studies): 12 months, baseline visit procedures will be used to confirm subject eligibility for this study
- For Group B (directly enrolled subjects): 12 months

Planned duration of safety follow-up:

- For Group A (subjects from antecedent studies): 7 days
- For Group B (directly enrolled subjects): 7 days

#### **Endpoints and statistical analysis:**

#### **Analysis Sets**

- Screened Set: all subjects who have provided informed consent.
- Enrolled Set: all subjects who have been assigned a subject identification number.
- <u>Safety Set</u>: all enrolled subjects who have taken at least 1 dose of study drug.
- <u>Full Analysis Set (FAS)</u>: all subjects in the safety set who completed at least 1 postdose efficacy assessment using ADHD-RS-5 Total score.

#### **Safety Endpoints**

Safety assessments include the occurrence of TEAEs and evaluations of blood pressure, pulse, weight, height, BMI; results of clinical laboratory, ECG, and sleep questionnaires (PSQ and CSHQ).

Additionally, the C-SSRS scale will capture the safety of SHP465 related to suicidality.

#### **Efficacy Endpoints**

The efficacy endpoint is defined as the change from baseline in the clinician-administered ADHD-RS-5 Total score.

The CGI-I will be a second efficacy and used to determine the proportion of subjects with an "improved" measurement based on the CGI-S measured at baseline. The CGI-I categories of "very much improved" and "much improved" will be classified as "improved" and all other assessed categories are grouped together as "not improved."

## **Statistical Methodology for Safety Endpoints**

Safety analyses will be summarized using the safety set, and presented by antecedent study treatment group and overall for TEAEs, clinical laboratory results, weight, height, BMI, vital signs, ECGs, PSQ, and CSHQ. The C-SSRS results will be summarized and listings of the C-SSRS data will be provided for subjects with a positive response.

## **Statistical Methodology for Efficacy Endpoints**

The FAS will be used to report the efficacy data. Descriptive summary statistics will be presented by antecedent study treatment group and overall for the observed efficacy variables. Change from baseline for the ADHD-RS-5 Total score at each on-therapy treatment visit will be summarized.

The number and proportion of subjects with an "improved" measurement in CGI-I will be reported at each applicable postdose visit. CGI-I scores will also be summarized.

# STUDY SCHEDULES

**Table 1: Schedule of Assessments for Group A** 

| Period | Baseline | | | | | | | Treatm | ent Peri | iod | | | | | | 1-Week Safety<br>Follow-up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit <sup>a</sup> | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16/ET <sup>b</sup> | Telephone<br>Call |
| Assessment<br>Week/Month | 0 | W1 | W2 | M1 | M2 | М3 | M4 | M5 | M6 | M7 | M8 | М9 | M10 | M11 | M12 | W53 |
| Assessment Day | 0 | 7 | 14 | 30 | 60 | 90 | 120 | 150 | 180 | 210 | 240 | 270 | 300 | 330 | 360 | 367 |
| Informed consent/assent | ✓ | | | | | | | | | | | | | | | |
| Inclusion/exclusion criteria <sup>c</sup> | ✓ | | | | | | | | | | | | | | | |
| Subject demographics | ✓ | | | | | | | | | | | | | | | |
| Medical and medication history <sup>d</sup> | ✓ | | | | | | | | | | | | | | | |
| Physical examination | ✓ | | | | | | | | | | | | | | ✓ | |
| Vital signs <sup>e, f</sup> | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | |
| Height <sup>g</sup> | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | |
| Weight <sup>g</sup> | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | |
| Clinical laboratory tests <sup>h</sup> | ✓ | | | | | | | | ✓ | | | | | | ✓ | |
| Electrocardiogram (12-lead) <sup>i</sup> | ✓ | | <b>√</b> | | ✓ | | ✓ | | ✓ | | ✓ | | ✓ | | ✓ | |
| Serum pregnancy test <sup>1</sup> | ✓ | | | | | | | | | | | | | | | |
| Urine pregnancy test <sup>1</sup> | | | | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | |
| ADHD-RS-5 <sup>k</sup> | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | |
| CGI-I <sup>j</sup> | | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | |
| PSQ <sup>j</sup> | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | |
| CSHQ <sup>j</sup> | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | |

**Table 1: Schedule of Assessments for Group A** 

| Period | Baseline | | Treatment Period | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit <sup>a</sup> | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16/ET <sup>b</sup> | Telephone<br>Call |
| Assessment<br>Week/Month | 0 | W1 | W2 | M1 | M2 | М3 | M4 | M5 | M6 | M7 | M8 | М9 | M10 | M11 | M12 | W53 |
| Assessment Day | 0 | 7 | 14 | 30 | 60 | 90 | 120 | 150 | 180 | 210 | 240 | 270 | 300 | 330 | 360 | 367 |
| C-SSRS Since Last<br>Visit version <sup>k</sup> | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | |
| Suitability of subject to remain in study <sup>j</sup> | ✓ | ✓ | ✓ | ✓ | <b>✓</b> | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | <b>√</b> | <b>✓</b> | | |
| Concomitant medications | ✓ | ✓ | <b>✓</b> | ✓ | <b>✓</b> | ✓ | <b>√</b> | <b>√</b> | ✓ | ✓ | <b>√</b> | ✓ | ✓ | <b>✓</b> | ✓ | <b>✓</b> |
| Adverse Events | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ |
| Access IWRS | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | |
| Investigational product distributed | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | <b>√</b> | | |
| Investigational product returned | | <b>√</b> | <b>√</b> | <b>√</b> | <b>✓</b> | ✓ | ✓ | ✓ | ✓ | <b>√</b> | ✓ | ✓ | ✓ | ✓ | ✓ | |
| Investigational product compliance | | ✓ | ✓ | <b>✓</b> | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | |

ADHD-RS-5=Attention-deficit/Hyperactivity Disorder Rating Scale 5, Child, Home Version; BMI=body mass index; CGI-I=Clinician's Global Impression – Improvement; CGI-S=Clinician's Global Impression – Severity of Illness; CSHQ=Children's Sleep Habits Questionnaire; C-SSRS=Columbia-Suicide Severity Rating Scale; ECG=electrocardiogram; ET=early termination; IWRS=interactive web response system; M=month; MINI-KID=Mini International Neuropsychiatric Interview for Children and Adolescents; PSQ=Post Sleep Questionnaire; TEAEs=treatment-emergent adverse events; W=week.

a Visit windows are with respect to baseline (Visit 2): ±2 days for Visit 3-4 and ±5 days for Visit 5-16 during treatment period, and +2 days for the safety follow up telephone call.

<sup>&</sup>lt;sup>b</sup> Subjects who terminate early will undergo the evaluations listed for Visit 16.

<sup>&</sup>lt;sup>c</sup> Inclusion/exclusion criteria will be reviewed at baseline (Visit 2).

<sup>&</sup>lt;sup>d</sup> Medical history will include all lifetime psychiatric and nonpsychiatric medications and procedures.

e Vital signs include oral or tympanic temperature, pulse, sitting blood pressure, and respiratory rate. The subject will have been seated for a minimum of 3 minutes before blood pressure, pulse, and respiratory rate measurements are taken. Measurement of blood pressure and pulse will be collected 3 times (with at least 2 minutes in between each collection) using the provided age-appropriate cuff. The average of each set of 3 measurements will be used to determine continued participation in the study.

f Blood pressure and pulse rate will be measured at each study visit. Temperature and respiratory rate will be measured at baseline (Visit 2).

<sup>&</sup>lt;sup>g</sup> Height and weight will be measured without shoes and with light clothing using a stadiometer for height and calibrated scale for weight.

<sup>&</sup>lt;sup>h</sup> Clinical laboratory evaluations will include hematology, biochemistry, endocrinology, and urinalysis.

<sup>&</sup>lt;sup>1</sup> Electrocardiograms will be recorded in triplicate with at least 3 minutes in between each collection at baseline only.

**Table 1: Schedule of Assessments for Group A** 

| Period | Baseline | | Treatment Period | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit <sup>a</sup> | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16/ET <sup>b</sup> | Telephone<br>Call |
| Assessment<br>Week/Month | 0 | W1 | W2 | M1 | M2 | М3 | M4 | M5 | M6 | M7 | M8 | М9 | M10 | M11 | M12 | W53 |
| Assessment Day | 0 | 7 | 14 | 30 | 60 | 90 | 120 | 150 | 180 | 210 | 240 | 270 | 300 | 330 | 360 | 367 |

JWhenever possible, the same individual should complete/rate consistently the following scales and questionnaires as appropriate: ADHD-RS-5, CGI-I, and subject check to remain in the study; PSQ, and CSHQ. Include assessment of decreased appetite.

k C-SSRS Pediatric/Cognitively impaired "Since Last Visit" version is completed for all visits. The scale will be compared with the C-SSRS Pediatric/Cognitively impaired "Baseline" from the antecedent study.

<sup>&</sup>lt;sup>1</sup>For females of child-bearing potential only.

**Table 2:** Schedule of Assessments for Group B

| Period | Scree<br>Wasl | | Baseline | | | | | | 7 | Freatm | ent Pe | riod | | | | | | 1-Week<br>Safety<br>Follow-up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit Number <sup>b</sup> | 1 | Phone call | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16/ET <sup>c</sup> | Telephone<br>Call |
| Assessment<br>Week/Month | -5 to -1 | -1 | 0 | W1 | W2 | M1 | M2 | М3 | M4 | M5 | M6 | M7 | M8 | М9 | M10 | M11 | M12 | W53 |
| Assessment Day <sup>b</sup> | −32 to −3 | -7 | 0 | 7 | 14 | 30 | 60 | 90 | 120 | 150 | 180 | 210 | 240 | 270 | 300 | 330 | 360 | 367 |
| Informed consent/assent | ✓ | | | | | | | | | | | | | | | | | |
| Inclusion/exclusion criteria <sup>d</sup> | ✓ | ✓ | ✓ | | | | | | | | | | | | | | | |
| Subject<br>demographics | ✓ | | | | | | | | | | | | | | | | | |
| MINI-KID | ✓ | | | | | | | | | | | | | | | | | |
| Medical and<br>medication history<br>includes prior<br>medications and<br>procedures <sup>e</sup> | <b>~</b> | | | | | | | | | | | | | | | | | |
| Urine drug screen | ✓ | | ✓g | | | | | | | | | | | | | | | |
| Serum pregnancy<br>test <sup>i</sup> | ✓ | | ✓g | | | | | | | | | | | | | | | |
| Urine pregnancy test <sup>i</sup> | | | ✓ | | | <b>√</b> | <b>✓</b> | <b>✓</b> | <b>✓</b> | <b>✓</b> | <b>✓</b> | <b>✓</b> | <b>✓</b> | <b>✓</b> | ✓ | ✓ | <b>~</b> | |
| ADHD-RS-5 <sup>f</sup> | | | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | |
| CGI-S <sup>f</sup> | | | ✓ | | | | | | | | | | | | | | | |
| CGI-I <sup>f</sup> | | | | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | |
| Physical examination | ✓ | | √g | | | | | | | | | | | | | | <b>✓</b> | |
| Height <sup>h</sup> | ✓ | | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | |
| Weight <sup>h</sup> | ✓ | | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | |
| Vital signs <sup>j, k</sup> | ✓ | | ✓g | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | |
| Clinical laboratory tests <sup>1</sup> | ✓ | | ✓g | | | | | | | | ✓ | | | | | | ✓ | |

**Table 2:** Schedule of Assessments for Group B

| Period | Scree<br>Wasl | | Baseline | | | | | | 7 | Freatm | ent Pe | riod | | | | | | 1-Week<br>Safety<br>Follow-up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit Number <sup>b</sup> | 1 | Phone call | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16/ET <sup>c</sup> | Telephone<br>Call |
| Assessment<br>Week/Month | -5 to -1 | -1 | 0 | W1 | W2 | M1 | M2 | М3 | M4 | М5 | M6 | M7 | M8 | М9 | M10 | M11 | M12 | W53 |
| Assessment Day <sup>b</sup> | −32 to −3 | -7 | 0 | 7 | 14 | 30 | 60 | 90 | 120 | 150 | 180 | 210 | 240 | 270 | 300 | 330 | 360 | 367 |
| Electrocardiogram (12-lead) <sup>m</sup> | ✓m | | <b>√</b> g, m | | ✓ | | ✓ | | ✓ | | ✓ | | ✓ | | ✓ | | ✓ | |
| C-SSRS baseline version <sup>f</sup> | ✓ | | | | | | | | | | | | | | | | | |
| C-SSRS since last<br>visit version <sup>f</sup> | | | <b>✓</b> | ✓ | ✓ | <b>✓</b> | ✓ | <b>✓</b> | <b>✓</b> | ✓ | ✓ | ✓ | <b>√</b> | <b>√</b> | ✓ | ✓ | ✓ | |
| PSQ <sup>f</sup> | | | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | |
| CSHQ <sup>f</sup> | | | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | |
| Adverse Events | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ |
| Concomitant medications | ✓ | ✓ | <b>✓</b> | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | <b>√</b> | ✓ | ✓ | ✓ | ✓ | ✓ |
| Suitability of<br>subject to remain<br>in study <sup>f</sup> | | | <b>√</b> | <b>√</b> | <b>✓</b> | <b>~</b> | <b>√</b> | <b>~</b> | <b>~</b> | ~ | ~ | <b>✓</b> | <b>√</b> | <b>√</b> | <b>√</b> | <b>√</b> | | |
| IWRS | ✓ | | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | |
| Study drug<br>dispensed | | | ✓ | ✓ | ✓ | <b>✓</b> | ✓ | <b>✓</b> | <b>✓</b> | <b>✓</b> | ✓ | ✓ | <b>✓</b> | ✓ | ✓ | ✓ | | |
| Study drug capsules returned | 1.6 | | Di 1 Di | ✓ | ✓ | ✓ | <b>✓</b> | ✓<br> | <b>✓</b> | ✓ | <b>✓</b> | <b>√</b> | <b>√</b> | <b>√</b> | ✓ | ✓ | ✓ | |

ADHD-RS-5 = Attention-deficit/Hyperactivity Disorder-Rating Scale 5, Child, Home Version; BMI=body mass index; CGI-I=Clinician's Global Impressions – Improvement; CGI-S=Clinician's Global Impressions – Severity of Illness; CSHQ=Children's Sleep Habits Questionnaire; C-SSRS=Columbia-Suicide Severity Rating Scale; ECG=electrocardiogram; ET=early termination; IWRS=interactive web response system; M=month; MINI-KID=Mini International Neuropsychiatric Interview for Children and Adolescents; PSQ=Post Sleep Questionnaire; W=week.

<sup>&</sup>lt;sup>a</sup> Following successful screening, a site representative will contact the subject's parent/LAR to instruct the subject on discontinuing any prohibited medication for the washout period.

b Visit windows are with respect to baseline (Visit 2): ±2 days for Visit 3-4 and ±5 days for Visit 5-16 during treatment period, and +2 days for the safety follow-up telephone call.

<sup>&</sup>lt;sup>c</sup> Subjects who terminate early will undergo the evaluations listed for Visit 16.

<sup>&</sup>lt;sup>d</sup> Inclusion/exclusion criteria will be reviewed during the washout telephone call and at baseline (Visit 2).

**Table 2: Schedule of Assessments for Group B** 

| Period | Scree<br>Wasl | 0 | Baseline | | Treatment Period | | | | | | | | | 1-Week<br>Safety<br>Follow-up | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit Number <sup>b</sup> | 1 | Phone call | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16/ET <sup>c</sup> | Telephone<br>Call |
| Assessment<br>Week/Month | -5 to -1 | -1 | 0 | W1 | W2 | M1 | M2 | М3 | M4 | M5 | M6 | M7 | M8 | М9 | M10 | M11 | M12 | W53 |
| Assessment Day <sup>b</sup> | −32 to −3 | -7 | 0 | 7 | 14 | 30 | 60 | 90 | 120 | 150 | 180 | 210 | 240 | 270 | 300 | 330 | 360 | 367 |

<sup>&</sup>lt;sup>e</sup> Medical history will include all lifetime psychiatric and nonpsychiatric medications and procedures.

<sup>&</sup>lt;sup>f</sup> Whenever possible, the same individual should complete/rate consistently the following scales and questionnaires as appropriate: ADHD-RS-5, CGI-S/I, and subject check to remain in the study; PSQ and CSHQ. Include assessment of decreased appetite.

g If >32 days have elapsed since the screening evaluation was completed at Visit 1, then the following evaluations must be repeated at baseline (Visit 2): vital signs, clinical laboratory evaluations, and ECGs in triplicate. The physical examination will be abbreviated with a review of the following body systems: general appearance, respiratory, and cardiovascular.

<sup>&</sup>lt;sup>h</sup> Height and weight will be measured without shoes and with light clothing using a stadiometer for height and calibrated scale for weight.

<sup>&</sup>lt;sup>i</sup> For females of child-bearing potential only

<sup>&</sup>lt;sup>j</sup> Vital signs include oral or tympanic temperature, pulse, sitting blood pressure, and respiratory rate. The subject will have been seated for a minimum of 3 minutes before blood pressure, pulse, and respiratory rate measurements are taken. Measurement of blood pressure and pulse will be collected 3 times (with at least 2 minutes in between each collection) using the age-appropriate cuff.

<sup>&</sup>lt;sup>k</sup> Blood pressure and pulse rate will be measured at each study visit. Temperature and respiratory rate will be measured at screening (Visit 1) only.

<sup>&</sup>lt;sup>1</sup> Clinical laboratory evaluations will include hematology, biochemistry, endocrinology, and urinalysis.

<sup>&</sup>lt;sup>m</sup> ECGs will be recorded in triplicate with at least 3 minutes in between each collection at screening only and at baseline only if >32 days have elapsed since the screening evaluation was completed at Visit 1.

#### 1 BACKGROUND INFORMATION

SHP465 extended-release capsules contain mixed salts of a single-entity amphetamine, a central nervous system (CNS) stimulant. The product was previously referred to as SPD465 however it is now being studied under the code of SHP465. SHP465 contains equal amounts (by weight) of 4 salts: dextroamphetamine sulfate and amphetamine sulfate, dextroamphetamine saccharate and amphetamine aspartate monohydrate. This results in a 3:1 mixture of dextro- to levo- amphetamine base equivalent.

SHP465 capsules are for oral administration. They contain 3 types of drug-releasing beads, an immediate release and 2 different types of delayed release (DR) beads. The first DR bead releases amphetamine at pH 5.5 and the other DR bead releases amphetamine at pH 7.0.

Amphetamines are noncatecholamine sympathomimetic amines with central nervous system stimulant activity. Amphetamine increases the availability of biogenic amines (primarily dopamine and norepinephrine) in central nerve terminals through multiple actions, including stimulating neurotransmitter release into the nerve terminal and inhibiting reuptake from the synapse. These actions may be the basis of its therapeutic actions in attention-deficit/hyperactivity disorder (ADHD); however, the mode of therapeutic action in ADHD is not known.

## 1.1 Indication and Current Treatment Options

The exact etiology of ADHD is unknown. Extensive research has suggested that neurotransmitter deficits (Arnsten, 2001), genetics (Arnsten, 2001; Brown, 2003), environment (Kahn et al., 2003), and perinatal complications (Bhutta and Anand, 2002) may all be contributing factors. The hypothesized mechanism of action of effective medications in ADHD is to raise neurotransmitter levels (specifically norepinephrine and/or dopamine, or their precursors) at the synapse either by facilitating neurotransmitter release from the synapse or by decreasing neurotransmitter reuptake by binding or activating the postsynaptic receptor (Kratochvil et al., 2003; Wang et al., 2007).

According to the Diagnostic and Statistical Manual of Mental Disorders, 5<sup>th</sup> edition (DSM-5), ADHD has 3 subtypes: hyperactive/impulsive, inattentive, and combined and individuals with ADHD may manifest considerably different symptomology depending on sex, disorder subtype, and the presence of comorbid disorders.

Compared with nonstimulants, stimulant medications (ie, amphetamine or methylphenidate) produce the most robust improvements in symptom expression across all age ranges (Spencer et al., 2001). Furthermore, stimulant medications have a rapid onset of action, within 1 to 2 hours of dosing, compared with nonstimulants (eg, atomoxetine), which can require dosing for up to 4 to 6 weeks to achieve maximal therapeutic benefit (Wilens et al., 2002).

Nonpharmacological measures (psychological, educational, and social) can also be beneficial and psychosocial treatments for adults with ADHD have been studied (Safren et al., 2004; Greenfield and Hechman, 2005).

Comorbid psychiatric and learning disorders are common in adults with ADHD and appropriate evaluation, diagnosis, and treatment are recommended (Weiss and Murray, 2003).

Importantly, symptoms may not only manifest throughout the day. Many patients continue to have residual symptoms lasting into the evening hours (Greenfield and Hechman, 2005). Adult patients may benefit from symptom relief into the evening hours for such activities as planning and organizing, or professional activities (eg, professional work at night), spousal/parental responsibilities, and driving. Similarly, impairments in nighttime activities are recognized in the pediatric population, which may need coverage all day and into the evening as well (eg, to do homework and to participate in family/social activities).

The impairments in psychosocial academic and occupational functioning associated with ADHD may arise from underlying chronic deficiencies in executive function (Brown, 1996). In general, the term executive function is used to describe a set of cognitive abilities that control and regulate judgments and behaviors which are necessary for goal-directed behavior; however, the specific definition of executive functioning varies and is debated. Understanding and treating executive functioning deficits is increasingly considered an unmet medical need in ADHD.

## 1.2 Product Background and Clinical Information

SHP465 and its prototypes have been evaluated in 1641 subjects in 16 clinical studies, of which 13 clinical studies were in adult subjects aged 18 to 55 years and 3 clinical studies were in pediatric subjects aged 6 to 17 years. The SHP465 clinical development program has shown that doses of 12.5 to 50 mg in adult subjects and 12.5 to 25 mg in pediatric subjects demonstrate a safety and efficacy comparable to the profile reflected in class labeling for stimulant products approved in the United States (US).

The pharmacokinetic (PK) profile of SHP465 is not affected if the capsule is consumed intact or if capsule contents are sprinkled onto a small amount of food (ie, 1 tablespoon of applesauce) and then ingested. The PK properties of SHP465 are not affected by sex or race. The PK properties between *d*- and *l*-amphetamine are similar.

Acceptable safety and tolerability profiles observed were consistent with the types of side effect specified in stimulant class labeling in the US. Specifically, administration of SHP465 was associated with increases in blood pressure (mean increase approximately 2-4 mmHg) and heart rate (mean increase approximately 3-6 bpm), and treatment-emergent adverse events (TEAEs) of insomnia, decreased appetite, decreased weight, heart rate increased, and anxiety, as well as psychiatric events (eg, mania, suicidality).

Always refer to the latest version of the SHP465 Investigator's Brochure (IB) for the overall risk/benefit assessment and the most accurate and current information regarding the drug metabolism, PK, efficacy, and safety of SHP465.

#### 2 STUDY OBJECTIVES AND PURPOSE

## 2.1 Rationale for the Study

The purpose of the study is to evaluate the long-term safety of SHP465 at 6.25 mg in children aged 4 to 12 years diagnosed with ADHD. Results from this study will provide important information on the long-term safety, tolerability, and efficacy of SHP465 at lower doses in the preschool/pediatric ADHD population.

## 2.2 Study Objectives

### 2.2.1 Primary Objective

The primary objective of this study is to evaluate the long-term safety and tolerability of SHP465 at 6.25 mg administered as a daily morning dose in children aged 4-12 years (inclusive at the time of consent) diagnosed with ADHD.

The evaluation of safety and tolerability will be based on the occurrence of treatment-emergent adverse events (TEAEs), evaluation of vital signs (systolic and diastolic blood pressure and pulse), weight, height, body mass index (BMI); clinical laboratory and electrocardiogram (ECG) results; sleep assessment (Post Sleep Questionnaire [PSQ], and Children's Sleep Habits Questionnaire [CSHQ]); and responses to the Columbia-Suicide Severity Rating Scale (C-SSRS).

## 2.2.2 Secondary Objectives

The secondary objectives of this study are as follows:

- 1. To describe the long-term efficacy of SHP465 using the clinician-administered ADHD Rating Scale 5 (ADHD-RS-5) Child, Home Version.
- 2. To describe the long-term efficacy of SHP465 using the Clinical Global Impressions-Improvement (CGI-I) scale.

IDENTIAL Page 26

18 May 2018

#### 3 STUDY DESIGN

## 3.1 Study Design and Flow Chart

This study is a Phase 3, long-term, open-label, multicenter, safety, and tolerability study in children (aged 4-12 years, inclusive, at the time of consent was obtained in the antecedent study [SHP465-112 or SHP465-309] or at the time of consent into this study if directly enrolled) with ADHD.

Approximately 145 subjects will be enrolled into this study. Subjects enrolled in this study will be divided into 2 groups based on participation in antecedent studies as follows:

- Subjects in Group A are those who have been rolled-over from antecedent studies (SHP465-112 or SHP465-309). These subjects do not need additional screening and washout procedures.
- Subjects in Group B will be directly enrolled subjects who will be required to undergo full screening and washout before enrollment.

Subjects in Group A will participate in the following 2 study periods: (1) treatment period and (2) safety follow-up. Subjects in Group B will participate in the following 3 study periods: (1) screening and washout, (2) treatment period, and (3) safety follow up.

For subjects in Group A, the last visit of the antecedent study, SHP465-112 or SHP465-309, will serve as the baseline visit (Visit 2) for this study. For subjects in Group B, a screening visit will precede a washout period.

The investigator or designee must obtain written informed consent from the subjects, if applicable, and the subject's parent/legally authorized representative (LAR) before any protocol-related procedure is performed. Procedures performed at each visit for all subjects are defined in the Study Schedules.

Figure 1: Study Design Flow Chart for Group A



Figure 2: Study Design Flow Chart for Group B



## 3.2 Duration and Study Completion Definition

Each subject's maximum duration of participation is expected to be approximately 12 months. The study will be completed in approximately 18 months.

Planned duration of screening/washout:

- For Group A (subjects from antecedent studies): None
- For Group B (directly enrolled subjects): up to 32 days

Planned duration of treatment:

- For Group A (subjects from antecedent studies): 12 months, baseline visit procedures will be used to confirm subject eligibility for this study
- For Group B (directly enrolled subjects): 12 months

Planned duration of safety follow-up:

- For Group A (subjects from antecedent studies): 7 days
- For Group B (directly enrolled subjects): 7 days

The study completion date is defined as the date the final subject, across all sites, completes their final protocol-defined assessment. Please note that this includes the follow-up visit or contact, whichever is later. The study completion date is used to ascertain timing for study results posting and reporting.

Subjects in both age groups will be treated and evaluated for 12 months and visit the site up to 15 times for subjects in Group A and up to 16 times for subjects in Group B.

## 3.3 Sites and Regions

The study will be conducted in approximately 50 sites in the US.


18 May 2018

#### 4 STUDY POPULATION

Each subject must participate in the informed consent process and provide written informed consent/assent before any procedures specified in the protocol are performed.

#### 4.1 **Inclusion Criteria**

The subject will not be considered eligible for the study without meeting all of the following criteria (including test results):

- 1. Subject is male or female aged 4 to 12 years, inclusive, at the time of consent for antecedent SHP465 trials (SHP465-112 or SHP465-309) in the ADHD population or at the time of consent for directly enrolled subjects into this study.
- 2. Subject's parent or legally authorized representative (LAR) must provide signature of informed consent, and there must be documentation of assent (if applicable) by the subject in accordance with the International Council on Harmonization (ICH) Good Clinical Practice (GCP) Guideline E6 (1996) and any updates and applicable regulations, before completing any study-related procedures.
- 3. Subject and parent/LAR are willing and able to comply with all of the testing and requirements defined in the protocol, including oversight of morning dosing. Specifically, the same parent/LAR should be available daily to dispense the dose of investigational product for the duration of the study.
- 4. For subjects in Group A:
  - Subject enrolled in the antecedent study SHP465-112 must have completed the treatment period and the pharmacokinetic (PK) sample collection (at the dose of 6.25 mg) without incidence of a clinically significant TEAE.
  - Subject enrolled in the antecedent study SHP465-309 must have completed the treatment period without reporting a clinically significant TEAE that would preclude subsequent exposure to SHP465.
- 5. For subjects in Group B (directly enrolled subjects), the following criteria must be met:
  - Subject meets the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for a primary diagnosis of ADHD (any subtype) based on a detailed psychiatric evaluation using the Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-KID)
  - Subject aged 4 to 5 years has an ADHD-RS-5 Child Version Total score of  $\geq$ 28 (boys) or  $\geq$ 24 (girls) at baseline (Visit 2)
  - Subject aged 6 to 12 years has an ADHD-RS-5 Child Version Total score of ≥28 at baseline (Visit 2)
  - Subject has a Clinical Global Impression–Severity of Illness score (CGI-S) ≥4 at baseline (Visit 2)
  - Subject has previously undergone an adequate course of nonpharmacological


18 May 2018

- treatment based on investigator judgment (aged 4-5 year olds) OR the subject is not completely satisfied with current adequate course of ADHD therapy (aged 6-12 year olds), OR the subject has a severe enough condition to consider enrollment without undergoing prior nonpharmacological treatment, based on investigator judgment.
- Subject functions as an age-appropriate level intellectually, based on investigator judgment.
- 6. Subject who is a female and of child-bearing potential must not have a positive serum beta human chorionic gonadotropin pregnancy test at the screening visit (Visit 1) and must have a negative urine pregnancy test at the baseline visit (Visit 2) and agree to comply with any applicable contraceptive requirements of the protocol.
- 7. Subject has lived with the same parent/LAR for at least 6 months.

#### 4.2 Exclusion Criteria

Subjects will be excluded from the study if any of the following exclusion criteria are met at baseline (Visit 2) for Group A or at screening (Visit 1) and/or baseline (Visit 2) for Group B.

These criteria apply to all subjects regardless of participation in an antecedent trial:

- 1. Subject was terminated from an antecedent SHP465 trial for noncompliance and/or had a serious TEAE during any previous SHP465 trial.
- 2. Subject is required to or is anticipated to take any medication that has central nervous system effects or affects performance, such as sedating antihistamines and decongestant sympathomimetics, or is a monoamine oxidase inhibitor. Stable use of bronchodilator inhalers is not exclusionary.
- 3. Subject has a concurrent chronic or acute illness (such as severe allergic rhinitis or an infectious process requiring antibiotics), disability, or other condition that might confound the results of safety assessments conducted in the study or that might increase risk to the subject. Similarly, the subject will be excluded if he or she has any additional condition(s) that, in the investigator's opinion, would prohibit the subject from completing the study or would not be in the best interest of the subject. The additional condition(s) would include any significant illness or unstable medical condition that could lead to difficulty complying with the protocol. Mild, stable asthma is not exclusionary.
- 4. Subject has a documented allergy, hypersensitivity, or intolerance to amphetamine or to any excipients in the investigational product.
- 5. Subject has a known family history of sudden cardiac death or ventricular arrhythmia.
- 6. Subject has a blood pressure measurement ≥95th percentile for age, sex, and height at screening (Visit 1) and/or baseline (Visit 2).
- 7. Subject has a height ≤5th percentile for age and sex at screening (Visit 1) and/or baseline (Visit 2).

- 8. Subject has a weight ≤5th percentile for age and sex at screening (Visit 1) and/or baseline (Visit 2).
- 9. Subject has a known history of symptomatic cardiovascular disease, structural cardiac abnormality, cardiomyopathy, serious heart rhythm abnormalities, or other serious cardiac conditions placing them at increased vulnerability to the sympathomimetic effects of a stimulant drug.
- 10. Subject has a history of seizures (other than infantile febrile seizures).
- 11. Subject has failed to fully respond, based on investigator judgment, to an adequate course of amphetamine therapy.
- 12. Subject is taking any medication that is excluded per the protocol.
- 13. Subject had any clinically significant ECG or clinical laboratory abnormalities at the screening (Visit 1) and/or baseline visit (Visit 2).
- 14. Subject has current abnormal thyroid function, defined as abnormal thyroid-stimulating hormone and thyroxine at the screening (Visit 1) and/or baseline visit (Visit 2). Treatment with a stable dose of thyroid medication for at least 3 months is permitted.
- 15. Subject has a current, controlled (requiring medication or therapy) or uncontrolled, comorbid psychiatric disorder including, but not limited to, any of the following comorbid Axis I disorders and Axis II disorders:
  - Post-traumatic stress disorder or adjustment disorder
  - Bipolar disorder, psychosis, schizophrenia or family history of these disorders
  - Pervasive developmental disorder
  - Obsessive-compulsive disorder
  - Serious tic disorder, or a family history of Tourette disorder
  - Any other disorder that in the opinion of the investigator contraindicates SHP465 or amphetamine treatment or confounds efficacy or safety assessments
- 16. Subject has a primary sleep disorder (eg., sleep apnea, narcolepsy)
- 17. Subject has a history or is currently diagnosed with an eating disorder
- 18. Subject is currently considered a suicide risk in the opinion of the investigator, has previously made a suicide attempt, or has a prior history of or currently demonstrating suicidal ideation.
- 19. Subject has a history of physical, sexual, or emotional abuse.
- 20. Subject has initiated behavioral therapy within 1 month before baseline (Visit 2). Subject may not initiate behavioral therapy during the study.
- 21. Subject has a clinically important abnormality on the urine drug and alcohol screen (except for the subject's current ADHD stimulant, if applicable) at screening (Visit 1) or baseline (Visit 2).
- 22. Subject is female and pregnant or lactating.
- 23. Subject cannot swallow a pill and/or applesauce or has an allergy to applesauce.

## **4.2.1** Female Contraception

Sexually active females of childbearing potential should be using an acceptable form of contraception. Females of childbearing potential must be advised to use acceptable contraceptives throughout the study period and for 30 days following the last dose of IMP. If hormonal contraceptives are used they should be administered according to the package insert. Females of childbearing potential who are not currently sexually active must agree to use acceptable contraception, as defined below, if they become sexually active during the period of the study and 30 days following the last dose of IMP.

Female children and adolescent subjects should be either:

- Premenarchal and either Tanner Stage 1 or <9 years, or
- Females of childbearing potential with a negative urine and/or serum beta-human chorionic gonadotropin (β-hCG) pregnancy test at screening and/or baseline (Group A and Group B subjects) and a negative urine pregnancy test at the baseline visit (Visit 2). Females of childbearing potential must agree to abstain from sexual activity that could result in pregnancy or agree to use acceptable methods of contraception.

Acceptable methods of contraception are:

- Intrauterine devices plus condoms
- Double-barrier methods (eg, condoms and diaphragms with spermicidal gel or foam)
- Hormonal contraceptives (oral, depot, patch, injectable, or vaginal ring), stabilized for ≥30 days before screening, plus condoms. Note: If subject becomes sexually active during the study, they should use 1 of the other acceptable methods noted above in addition to the hormonal contraceptive until it has been stabilized for 30 days.

## 4.2.2 Male Contraception

Male subjects must agree to either abstain from sex or to use condoms if they become sexually active during the period of the study and for 30 days following the last dose of investigational product.

## 4.3 Discontinuation of Subjects

A subject may withdraw from the study, or the parent/LAR may withdraw the subject from the study, at any time for any reason without prejudice to their future medical care by the physician or at the institution. The investigator or sponsor may withdraw the subject at any time (eg, in the interest of subject safety). The investigator is encouraged to discuss withdrawal of a subject from investigational product with the medical monitor when possible.

If investigational product is discontinued, regardless of the reason, the evaluations listed for Visit 16/early termination (ET) are to be performed as completely as possible. Whenever possible, all discontinued subjects should also undergo the protocol-specified follow-up. Comments (spontaneous or elicited) or complaints made by the subject must be recorded in the

FIDENTIAL Page 32

18 May 2018

source documents. The reason for termination, date of stopping investigational product, and the total amount of investigational product taken must also be recorded in the source documents and the most clinically relevant reason should be entered on the CRF.

Subjects who discontinue will not be replaced.

## 4.3.1 Management of Blood Pressure and Pulse During the Study

To ensure that potential blood pressure and pulse increases associated with the use of SHP465 in this population are carefully monitored and appropriately managed, all subjects must be further evaluated if they meet any of the criteria defined in Sections 4.3.1.1 and 4.3.1.2.

## 4.3.1.1 Systolic and Diastolic Blood Pressure

Blood pressure criteria for further evaluation have been developed based on the normative data presented in the National Institutes of Health Fourth Report on the Diagnosis, Evaluation, and Treatment of High Blood Pressure in Children and Adolescents (NIH, 2004).

Prior to obtaining vital signs (blood pressure and pulse) the subjects should be at rest for at least 3 minutes.

If any subject's blood pressure measurements meet either criterion below, the investigator will notify the medical monitor. If any subject's blood pressure measurements meet either criterion below on 3 consecutive visits, the subject should be considered for potential discontinuation based upon the clinical judgment of the investigator and in conjunction with the medical monitor

- Elevations in the average (of 3 readings) sitting systolic blood pressure defined as an increase of >15 mmHg from the baseline visit (Visit 2) OR a value >95th percentile for age, sex, and height.
- Elevations in average (of 3 readings) sitting diastolic blood pressure defined as an increase of >15 mmHg from the baseline visit (Visit 2) OR an average (of 3 readings) sitting diastolic blood pressure value >95th percentile for age, sex, and height.

Any subject with a systolic or diastolic blood pressure measurement <95<sup>th</sup> percentile for age, sex, and height percentile may be discontinued from the study based upon the clinical judgment of the investigator regarding the subject's safety.

#### 4.3.1.2 Pulse

The resting pulse rate criterion for further evaluation has been defined based on the normative data presented in the National Health Statistics Report's "Resting Pulse Rate Reference Data for Children, Adolescents, and Adults: United States, 1999-2008" (Ostchega et al., 2011).

Any subject that has a resting, sitting pulse rate >126 bpm for age 4-5 years or >116 bpm for age 6-12 years based on the average of 3 readings or is symptomatic requires further assessment. In this case an unscheduled visit needs to be conducted within 1 business day. At the unscheduled visit, if the subject's pulse rate remains above the criteria based on the average of 3 readings or if

SHP465-308

18 May 2018

the subject is symptomatic then the subject's investigator will discuss the findings with the medical monitor. In careful consideration of the subject's pulse value, magnitude of increase from baseline and symptoms, a joint decision between the investigator and the medical monitor will be made regarding continued participation in the study. If a visit cannot be scheduled the next day, the subject may be discontinued from the study.

Any subject with a pulse rate equal or lower than the number for age defined above may be discontinued from the study based upon the clinical judgment of the investigator regarding the subject's safety.

#### 4.3.2 Reasons for Discontinuation

The reason for withdrawal must be determined by the investigator and recorded in the subject's medical record and source documents. If a subject is withdrawn for more than 1 reason, each reason should be documented in the source documents.

Reasons for discontinuation include but are not limited to:

- Adverse event
- Protocol violation
- Withdrawal by subject or parent/LAR
- Lost to follow-up
- Lack of efficacy
- Blood pressure and/or pulse criteria met
- Other (must be specified)

## 4.3.3 Subjects "Lost to Follow-up" Prior to Last Scheduled Visit

A minimum of 3 documented attempts must be made to contact the parent/LAR of any subject lost to follow-up at any time point before the last scheduled contact (office visit or telephone contact). At least 1 of these documented attempts must include a written communication sent to the subject's last known address via courier or mail (with an acknowledgement of receipt request) asking that they return to the site for final safety evaluations and return any unused investigational product.

#### 5 PRIOR AND CONCOMITANT TREATMENT

#### **5.1** Prior Treatment

Prior treatment includes all treatment (including but not limited to herbal treatments, vitamins, behavioral treatment, nonpharmacological treatment such as psychotherapy) received within 30 days (or PK equivalent of 5 half-lives, whichever is longer) prior to the date of first dose of investigational product. Prior treatment information must be recorded in the subject's source documents.

Washout for all prior medications must be a minimum of 5 times the half-life of the medication.

#### **5.2** Concomitant Treatment

Concomitant treatment refers to all treatment taken between the dates of the first dose of investigational product and the end of the follow-up period, inclusive. Concomitant treatment information must be recorded in the appropriate source document.

#### **5.2.1** Permitted Treatment

Medications permitted during the study are listed as follows:

- Stable (ie, for at least 3 months before the baseline visit [Visit 2] for subjects in Group A and the screening/washout visit [Visit 1] for subjects in Group B) dose of thyroid medication is permitted
- Stable (ie, for at least 1 month before the baseline visit [Visit 2] for subjects in Group A and the screening/washout visit [Visit 1] for subjects in Group B) dose of bronchodilator inhalers (however, beta-agonists and chronic use of oral corticosteroids are prohibited)
- Any medications that do not affect blood pressure, heart rate, or the central nervous system, and which are considered necessary for the subject's welfare, may be administered at the discretion of the investigator
- Nonsedating antihistamines such as fexofenadine (eg, Allegra<sup>®</sup>, Sanofi), loratadine (eg, Claritin<sup>®</sup>, Schering-Plough), and cetirizine hydrochloride (eg, Zyrtec<sup>®</sup>, McNeil-PPC)
- Over-the-counter nonstimulant cold remedies

Concomitant psychotherapy must also be recorded in the appropriate section of the source documents.

### **5.2.2** Prohibited Treatment

Table 3 details the washout period, relative to the baseline visit (Visit 2), for treatments that are excluded during this study. Subjects can only be instructed to discontinue a medication for this study after informed consent has been obtained.

Table 3: Common Excluded Treatments and Associated Washout Period - Relative to Baseline Visit (Visit 2)

| | Nui | Minimumber of fore Base Visit | Days seline |
|---|---|---|---|
| Treatment | 7 | 14 | 30 |
| Psychostimulants, amphetamines, and amphetamine-like agents | X | | |
| Antihypertensives <sup>a</sup> | X | | |
| Antihistamines (centrally and peripherally active) | | X | |
| Herbal preparations (including melatonin) | | X | |
| Sedatives, anxiolytics, antipsychotics <sup>a</sup> | | | X |
| Monoamine oxidase inhibitors <sup>a</sup> | | | X |
| Antidepressants <sup>a</sup> | | | X |
| Clonidine and guanfacine | | | X |
| Selective noradrenaline reuptake inhibitors and noradrenaline reuptake inhibitors <sup>a</sup> | | | X |
| CYP2D6 inhibitors (eg, paroxetine, fluoxetine, quinidine, ritonavir) | | | X |
| Alkalinizing agents (eg, sodium bicarbonate, acetazolamide, some thiazides) | | | X |
| Acidifying agents (eg, guanethidine, reserpine, glutamic acid HCl, ascorbic acid, ammonium chloride, sodium acid phosphate, methenamine salts) | | | X |

<sup>&</sup>lt;sup>a</sup> These medications may signal that an exclusionary diagnosis is present. The medical monitor should be consulted before instructing a subject to discontinue 1 of these medications for this study.

FIDENTIAL Page 36

18 May 2018

#### 6 INVESTIGATIONAL PRODUCT

## 6.1 Identity of Investigational Product

The test product is SHP465, which will be provided in 6.25 mg capsule form. The product was previously referred to as SPD465 and is registered with the Drug Enforcement Agency (DEA) as SPD465; however, it is now being studied under the code of SHP465. The drug will be labeled with SHP465 (SPD465).

## **6.1.1** Blinding the Treatment Assignment

Not applicable.

## 6.2 Administration of Investigational Product(s)

## 6.2.1 Interactive Response Technology for Investigational Product Management

An interactive web response system (IWRS) will be employed in this study to manage the tracking and confirmation of shipments, supply, inventory, ordering, expiration, site assignments, and dosing of the investigational products.

The IWRS provider will provide a user manual and training to each site, with detailed instruction on the use of the IWRS.

## 6.2.2 Allocation of Subjects to Treatment

All subjects will receive open-label SHP465 during this study.

Subject numbers are assigned to all subjects as they consent to take part in the antecedent study or this study if directly enrolled. Within each site (numbered uniquely within a protocol), the subject number is assigned to subjects according to the sequence of presentation for study participation.

## **6.2.3 Dosing**

Dosing should begin at 7:00 AM ( $\pm 2$  hours) on the morning after the baseline visit (Visit 2). The parent/LAR responsible for dosing will be instructed to dispense 1 capsule to the subject daily in the morning throughout the study, at approximately the same time each day. The same parent/LAR should be available daily to dispense the dose of investigational product for the study duration.

SHP465 may be administered in 1 of the following ways:

- Swallow SHP465 capsule whole, or
- Open capsule and sprinkle the entire contents on applesauce

The sprinkled applesauce should be consumed immediately; it should not be stored. Subjects should take the sprinkled applesauce in its entirety without chewing. The dose of a single capsule should not be divided. The empty capsule shells should be discarded.
Subjects will be treated with SHP465 at 6.25 mg.

The investigator will categorize subject response into 1 of the following 3 conditions, along with the associated actions:

- <u>Intolerable response</u> (ie, subject experiences intolerable side effects): If this lower dose also produces an intolerable effect, the subject should be discontinued from the study.
- <u>Ineffective response</u> (ie, subject has not achieved at least a 30% reduction in ADHD-RS-5 Child, Home Version total score from the baseline visit [Visit 2] and a CGI-I score of 1 or 2).
- Acceptable response (ie, subject has achieved at least a 30% reduction in ADHD-RS-5 Child, Home Version total score from the baseline visit [Visit 2] and a CGI-I score of 1 or 2 with tolerable side effects): This response suggests that an optimal dose has been achieved and the subject should maintain this dose for the remainder of the study.

If the subject experiences unacceptable tolerability, in the opinion of the clinician, the subject will be discontinued.

# **6.2.4** Unblinding the Treatment Assignment

Not applicable.

### 6.3 Labeling, Packaging, Storage, and Handling

#### 6.3.1 Labeling

Labels containing study information and pack identification are applied to the investigational products container.

All investigational product is labeled with a minimum of the protocol number, medication identification number (if applicable), dosage form (including product name and quantity in pack), directions for use, storage conditions, expiry date (if applicable), batch number and/or packaging reference, the statement "CAUTION: New Drug - Limited by Federal (or United States) Law to Investigational Use", "Keep out of reach of children", and the sponsor's name and address. Any additional labeling requirements for participating countries and/or controlled substances will also be included on the label.

Space is allocated on the label so that the site representative can record a unique subject identifier and initials.

Additional labels (eg, those used when dispensing marketed product) may, on a case-by-case basis, be applied to the investigational product in order to satisfy local or institutional requirements, but must not:

• Contradict the clinical study label


- Obscure the clinical study label
- Identify the study subject by name

Additional labels may not be added without the sponsor's prior full agreement.

# 6.3.2 Packaging

Investigational product is packaged in the following labeled containers:

SHP465 capsules are packaged in 9-count high-density polyethylene bottles with child-resistant closures.

Changes to sponsor-supplied packaging before dosing may not occur without full agreement in advance by the sponsor.

# 6.3.3 Storage

The investigator has overall responsibility for ensuring that the investigational product is stored in a secure, limited-access location. Limited responsibility may be delegated to the pharmacy or member of the study team, but this delegation must be documented. Investigational products are distributed by the pharmacy or nominated member of the study team. The pharmacist/nominated team member will enter the unique subject identifier and initials on the investigational product bottle/carton labels as they are distributed.

Investigational product must be stored in accordance with labeled storage conditions. Temperature monitoring is required at the storage location to ensure that the investigational product is maintained within an established temperature range. The investigator is responsible for ensuring that the temperature is monitored throughout the duration of the study and that records are maintained; the temperature should be monitored continuously by using either an in-house system, a mechanical recording device such as a calibrated chart recorder, or by manual means, such that both minimum and maximum thermometric values over a specific time period can be recorded and retrieved as required. Such a device (ie, certified minimum/maximum thermometer) would require manual resetting upon each recording. The sponsor must be notified immediately upon discovery of any excursion from the established range. Temperature excursions will require site investigation as to cause and remediation. The sponsor will determine the ultimate impact of excursions on the investigational product and will provide supportive documentation as necessary. Under no circumstances should the product be dispensed to subjects until the impact has been determined and the product is deemed appropriate for use by the sponsor.

The sponsor should be notified immediately if there are any changes to the storage area of the investigational product that could affect the integrity of the product(s), eg, fumigation of a storage room.

All controlled-substance investigational product for the sponsor's studies must be stored in a securely locked, substantially constructed room or cabinet according to all applicable local, state, and/or national laws. Limited, controlled access to these investigational products must be maintained, as well as chain of custody, for all investigational product movement.

# 6.4 Drug Accountability

Investigators will be provided with sufficient amounts of the investigational product to carry out this protocol for the agreed number of subjects. The investigator or designee will acknowledge receipt of the investigational product, documenting shipment content and condition. Accurate records of all investigational product dispensed, used, returned, and/or destroyed must be maintained as detailed further in this section.

The investigator has the overall responsibility for administering/dispensing the investigational product. Where permissible, tasks may be delegated to a qualified designee (eg, a pharmacist) who is adequately trained in the protocol and who works under the direct supervision of the investigator. This delegation must be documented in the applicable study delegation of authority form. The investigator or designee will be required to have a valid DEA Form 223 certificate of registration for 2N Controlled Substances for the duration of the study and be able to order and distribute 2N Controlled Substances via a valid DEA Form 222.

The investigator or designee (as documented by the investigator in the applicable study delegation of authority form) will dispense the investigational product only to the parent/LAR of subjects included in this study following the procedures set out in the study protocol. The parent/LAR of each subject will be given only the investigational product carrying the subject's treatment assignment. All dispensed medication will be documented on the source documents and/or other investigational product record.

The investigator is responsible for ensuring the retrieval of all study supplies from each subject's parent/LAR.

No investigational product stock or returned inventory from a Shire-sponsored study may be removed from the site where originally shipped without prior knowledge and consent by the sponsor. If such transfer is authorized by the sponsor, all applicable local, state, and national laws must be adhered to for the transfer.

The sponsor or its representatives must be permitted access to review the supplies storage and distribution procedures and records.

At the end of the study, or as instructed by the sponsor, all unused stock, subject-returned investigational product, and empty/used investigational product packaging are to be sent to a nominated contractor on behalf of the sponsor. Investigational products being returned to the sponsor's designated contractors must be counted and verified by clinical site personnel and the sponsor (or designated contract research organization [CRO]). For unused supplies where the original supplied tamper-evident feature is verified as intact, the tamper-evident feature must not be broken and the labeled amount is to be documented in lieu of counting. Shipment return forms, when used, must be signed before shipment from the site. Validated electronic return systems (ie, interactive response technology) do not require a shipment form. Returned investigational products must be packed in a tamper-evident manner to ensure product integrity. Contact the sponsor for authorization to return any investigational product before shipment. Shipment of all returned investigational product must comply with local, state, and national laws. As this is a controlled substance, investigational product cannot be destroyed at site, and must be

returned to the depot. All DEA Form 222s will be required to accompany any site shipments and site returns back to the depot. Accountability must be performed at the capsule level.

Based on entries in the site drug accountability forms, it must be possible to reconcile investigational products delivered with those used and returned. All investigational products must be accounted for and all discrepancies investigated and documented to the sponsor's satisfaction.

# 6.5 Subject Compliance

The parent/LAR of each subject must be instructed to bring their unused investigational product and empty/used investigational product packaging to every visit. Drug accountability must be assessed at the container/packaging level for unused investigational product that is contained within the original tamper-evident sealed container (eg, bottles, trays, vials) or at the individual count level for opened containers/packaging. The pharmacist/nominated person will record details on the drug accountability form.

#### 7 STUDY PROCEDURES

# 7.1 Study Schedule

The schedules of assessments (Table 1 [Group A] and Table 2 [Group B]) detail all procedures to be completed at each visit and should serve as the primary section of the protocol regarding visit-specific study procedures.

Clinician-completed rating scales and assessments conducted by the site, ie, ADHD-RS-5, CGI-S, CGI-I, and C-SSRS must be completed by the same rater whenever possible. The parent/LAR completed PSQ and CSHQ should be completed by the same individual whenever possible.

For both groups throughout the treatment period, visits should be scheduled as outlined ( $\pm 2$  days for Visit 3-4 and  $\pm 5$  days for Visit 5-16), with reference to the baseline visit (Visit 2). The safety follow-up call should be scheduled 7 days after the final dose with a +2-day visit window.

For Group A, the subjects will be required to visit the site up to 15 times and for Group B, the subjects will be required to visit the site up to 16 times over a 12-month period.

Additional unscheduled visits and/or assessments may occur as needed for safety (eg, unscheduled visits for blood pressure and/or pulse measurements).

# 7.1.1 Screening and Washout Period (Group A and Group B)

For subjects in Group A, the last visit of the antecedent study, SHP465-112 or SHP465-309, will serve as the baseline visit (Visit 2) for this study. The investigator or designee must obtain written informed consent from the subject's parent/LAR prior to any procedures related to this protocol being performed.

Subjects in Group B are directly enrolled subjects and will be required to undergo full screening and washout before enrollment. A separate screening visit will be conducted followed by a washout period for subjects in Group B.

The principal investigator or designee must obtain written informed consent from the subject's parent/LAR before any SHP465-308 study-related procedures are conducted during the screening visit (Visit 1). There must also be documentation of assent (if required by the Institutional Review Board [IRB]), indicating that the subject is aware of the investigational nature of the study and the required procedures and restrictions, before the performance of any SHP465-308 study-related procedures.

A subject cannot be instructed to washout any medication for this study until after informed consent is obtained.

Screening procedures may take place across multiple days to allow enough time to complete all procedures and confirm initial subject eligibility. Screening procedures and dates should be well documented in the source documents. The date of the screening visit (Visit 1) is the date the subject and parent/LAR has signed informed consent for this study. Subjects requiring washout

must have an abbreviated physical examination, clinical laboratory tests, and 12-lead ECG repeated if >32 days have elapsed since the safety measurements at the screening visit (Visit 1) were collected.

# 7.1.1.1 Screening Visit (Visit 1) for Group B

Subjects in Group B will be screened at Visit 1 to establish eligibility for study participation.

Table 2 (Group B) details all procedures to be completed at the screening visit (Visit 1) and should serve as the primary point of reference regarding study procedures. Additional clarification on the procedures performed during the screening visit (Visit 1) is as follows:

- Eligibility will be established per inclusion and exclusion criteria, including documentation of any prior nonpharmacological treatment, specified MINI-KID, and C-SSRS criteria. Areas of impairment will be recorded for all subjects for assessing the severity of the subject's condition.
- All adverse events (AEs) occurring after signature of informed consent must be recorded in the source documents.
- Three 12-lead ECGs will be taken, with approximately 3 minutes in between each one, to ensure that appropriate baseline intervals are established. The investigator will perform the initial interpretation of the ECG immediately after collection to ensure the safety of each subject. The ECG tracing will be sent to the central reader for analysis. Upon review of the report from the central reader, the investigator will re-evaluate the clinical significance of the ECG in light of other safety data for the subject. If abnormal and significant results are observed following assessment by the central reader, the investigator, in consultation with the appointed CRO medical monitor, will confirm the subject's eligibility to participate in this study.
- Vitals will include oral or tympanic temperature, pulse, sitting blood pressure, and respiratory rate. Also, blood pressure and pulse will be collected 3 times (with at least 2 minutes in between each collection) using the age-appropriate cuff during the visit. The average of each set of 3 measurements will be used to determine continued participation in the study (see Section 4.3.1).
- Height and weight will be measured without shoes.
- The "baseline" version of the Pediatric/Cognitively Impaired Version C-SSRS should be completed.
- Clinical lab tests will include hematology, biochemistry, endocrinology, and urinalysis.
- Historical/concomitant medications will be recorded as follows:
  - All lifetime psychoactive medications and lifetime nonpharmacological interventions (behavioral therapy) for ADHD
  - Other medications used during the 30 days before the screening visit (Visit 1)


A screen failure is a subject who has given informed consent and failed to meet the inclusion and/or met at least 1 of the exclusion criteria and has not been randomized or administered investigational products. Subjects cannot be rescreened once they have been designated as a screen failure.

# 7.1.1.2 Washout Telephone Call (Group B)

The washout period will be initiated after clinical laboratory test results and 12-lead ECG results have been received and reviewed by the investigator.

Eligible subjects will be contacted by a member of the site staff and provided with instructions on discontinuing any protocol-prohibited medications. During washout, a subject's current prohibited medications (if applicable) will be discontinued for a period of up to 32 days or 5 times the half-life of the medication, whichever is longer. Washout periods for prohibited medications are defined in Table 3.

As part of the washout telephone call, site personnel will perform the following procedures:

- Schedule the baseline visit (Visit 2)
- Review the inclusion/exclusion criteria
- Ask about any concomitant medications that the subject is taking. If new concomitant
  medications that require washout are noted, instructions for appropriate washout will
  be provided
- Provide instructions on discontinuing any medication requiring washout
- Determine if any AEs have occurred since the screening visit (Visit 1)

If a medication washout is not necessary, the washout telephone call will include all the above procedures except providing instructions on discontinuing any current medications.

#### 7.1.1.3 Baseline Visit (Visit 2) Group A

Visit 2 for subjects in Group A will be the same day as the final on-site visit for the antecedent study. During this visit, subjects will be screened for eligibility into study SHP465-308.

The investigator or designee must obtain written informed consent from the subject's parent/LAR before any SHP465-308 study-related procedures conducted during the baseline visit (Visit 2). There must also be documentation of assent (if required by IRB), indicating that the subject is aware of the investigational nature of the study and the required procedures and restrictions, before the performance of any SHP465-308 study-related procedures.

Inclusion/exclusion criteria must be reviewed during this visit to ensure subjects continue to meet all eligibility criteria.

Table 1 (Group A) outlines all procedures to be conducted during Visit 2 and should serve as the primary point of reference regarding study procedures. Additional clarification on the procedures performed during the baseline visit (Visit 2) is provided as follows:


18 May 2018

- Vitals will include oral or tympanic temperature, pulse, sitting blood pressure, and respiratory rate. Also, blood pressure and pulse will be collected 3 times (with at least 2 minutes in between each collection) using the age-appropriate cuff during the visit. The average of each set of 3 measurements will be used to determine continued participation in the study (Section 4.3.1).
- For eligible subjects, the investigator or assigned site staff designee will access the IWRS to enroll the subject and obtain an investigational product bottle number to dispense to the subject's parent/LAR. Sufficient investigational product will be dispensed to last until the next regularly scheduled visit. The parent/LAR responsible for dosing will be instructed to dispense 1 capsule each day to the subject. Dosing will begin the morning after the baseline visit (Visit 2).
- The C-SSRS "Since Last Visit" Version of the Pediatric/Cognitively Impaired Version should be completed.

# 7.1.1.4 Baseline Visit (Visit 2) Group B

Once the screening central clinical laboratory tests and 12-lead ECG results have been obtained, in addition to repeat assessments (if required), and the subject has completed the required washout period (if applicable), the subject will return to the site for the baseline visit (Visit 2).

Inclusion/exclusion criteria must also be reviewed during this visit to ensure that the subject continues to meet all eligibility criteria.

Table 2 (Group B) outlines all procedures to be conducted during the baseline visit (Visit 2) and should serve as the primary point of reference regarding study procedures. Additional clarification on the procedures performed during the baseline visit (Visit 2) is provided as follows:

- For subjects with >32 days since the safety measurements at the screening visit (Visit 1) were collected, an abbreviated physical examination, vital signs, clinical laboratory tests, and 12-lead ECG in triplicate must be repeated, and the results reviewed by the investigator before the subject is enrolled.
- Blood pressure and pulse will be collected 3 times (with at least 2 minutes in between each collection) using the age-appropriate cuff during the visit. The average of each set of 3 measurements will be used to determine continued participation in the study (see Section 4.3.1).
- If >32 days since the screening visit (Visit 1), 3 ECGs will be taken, with approximately 3 minutes in between each one, to ensure that appropriate baseline intervals are established. The investigator will perform the initial interpretation of the ECG immediately after collection to ensure the safety of each subject to continue with the study. The ECG tracing will be sent to the central reader for analysis. Upon review of the report from the central reader, the investigator will re-evaluate the clinical significance of the ECG in light of other safety data for the subject. If abnormal and significant results are observed following assessment by the central reader, the investigator, in consultation with the appointed CRO medical monitor, will

- confirm the subject's continued participation in this study.
- The C-SSRS "Since Last Visit" Version of the Pediatric/Cognitively Impaired Version should be completed.
- For eligible subjects, the investigator or assigned site staff designee will access the IWRS to enroll the subject and obtain an investigational product bottle number to dispense to the subject's parent/LAR. Sufficient investigational product will be dispensed to last until the next regularly scheduled visit. The parent/LAR responsible for dosing will be instructed to dispense 1 capsule each day to the subject. Dosing will begin the morning after the baseline visit (Visit 2).

# 7.1.2 Treatment Period (Group A and Group B)

At each visit during the treatment period up to and including Visit 16, sufficient investigational product will be dispensed to last until the next regularly scheduled visit. The parent/LAR responsible for dosing will be instructed to dispense 1 capsule each day to the subject. At each visit, the subject's parent/LAR must return any empty or unused bottles to permit drug accountability and compliance to be assessed.

Throughout the treatment period, subjects may attend the clinic for unscheduled visits to address any medical needs that arise between scheduled visits.

Table 1 (Group A) and Table 2 (Group B) outline all procedures to be conducted during Visits 3 and 4 and should serve as the primary point of reference regarding study procedures. Further clarification for these visits is outlined as follows:

- At Visits 3 and 4, subjects must return any empty or unused bottles to permit drug accountability and compliance to be assessed.
- Subjects will be dispensed a 9-count bottle of investigational product to cover them until their next regularly scheduled visit. Subjects will be instructed to take 1 capsule each day. Dosing will begin the morning after each visit.
- Blood pressure and pulse will be collected 3 times (with at least 2 minutes in between each collection) using the age-appropriate cuff during the visit. The average of each set of 3 measurements will be used to determine continued participation in the study (see Section 4.3.1).
- Scales should be completed by the same rater with input from the same parent/LAR whenever possible.
- The C-SSRS "Since Last Visit" Version of the Pediatric/Cognitively Impaired Version should be completed during Visits 3 and 4.

### 7.1.2.1 Treatment Period (Visits 5 to 16/Early Termination)

Subjects will continue daily morning treatment for an additional 12 months.

Throughout the treatment period, subjects may attend the clinic for unscheduled visits to address any medical needs that arise between scheduled visits.

Table 1 (Group A) and Table 2 (Group B) outline the procedures to be completed at each visit during the treatment period and should serve as the primary point of reference regarding study procedures. Additional clarification on the procedures to be performed during the treatment period Visits 5 to 16 is provided as follows:

- Scales are to be completed by the same rater with input from the same parent/LAR whenever possible
- At each visit during the treatment period, subjects must return any empty or unused bottles to permit drug accountability and compliance to be assessed
- Subjects will be dispensed a 9-count bottle of investigational product to cover them until their next regularly scheduled visit. Subjects will be instructed to take 1 capsule each day. Dosing will begin the morning after each visit.
- The C-SSRS "Since Last Visit" Version of the Pediatric/Cognitively Impaired Version should be completed during the treatment period.
- Blood pressure and pulse will be collected 3 times (with at least 2 minutes in between each collection) using the age-appropriate cuff during the visit. The average of each set of 3 measurements will be used to determine continued participation in the study (see Section 4.3.1).

All subjects who complete the study or discontinue early will complete Visit 16/ET.

Table 1 (Group A) and Table 2 (Group B) outline all procedures to be conducted during Visit 16/ET and should serve as the primary point of reference regarding study procedures.

Further clarification on the procedures performed during Visit 16/ET is provided as follows:

- Unused investigational product and empty containers will be collected to calculate medication compliance.
- Blood pressure and pulse will be collected 3 times (with at least 2 minutes in between each collection) using the age-appropriate cuff during the visit. The average of each set of 3 measurements will be used to determine continued participation in the study (see Section 4.3.1).

### 7.1.3 Safety Follow-up Period (Group A and Group B)

The follow-up period for this protocol is 7 days (+2 days) from the final dose of investigational product.

At the end of this period, there will be a telephone call initiated by the site staff to query for serious adverse events (SAEs), TEAEs, and concomitant treatments. All TEAEs and SAEs that are not resolved at the time of this contact will be followed to closure (see Section 8.1).

SHP465-308

18 May 2018

# 7.1.4 Additional Care of Subjects After the Study

No aftercare is planned for this study. The investigator will discuss the available ADHD treatment options for subjects.

# 7.2 Study Evaluations and Procedures

The individual indicated in each scale description will perform all assessments listed as follows. Assessments are to be performed according to the schedule shown in Table 1 (Group A) and Table 2 (Group B). Care must be taken by the site personnel or the investigator to fully explain the scale before completion.

If the subject terminates treatment early, all assessments listed in Table 1 (Group A) and Table 2 (Group B) for Visit 16/ET and the safety follow-up call should be completed. Whenever possible, raters (including parent/LAR, and the investigator or site designee) observing the subject's behavior should be consistent from visit to visit throughout the study.

# 7.2.1 Demographic and Other Baseline Characteristics

Demographic characteristics such as age, sex, weight, height, and BMI will be collected throughout the study according to Table 1 (Group A) and Table 2 (Group B).

# 7.2.1.1 Mini International Neuropsychiatric Interview for Children and Adolescents

The MINI-KID is a structured clinical diagnostic interview designed to assess the presence of psychiatric disorders in children and adolescents in a way that is comprehensive and concise. It follows the structure and format of the adult version of the interview and is organized in diagnostic sections or modules. Using branching tree logic, the instrument asks 2 to 4 screening questions for each disorder. Additional symptom questions within each disorder section are asked only if the screen questions are positively endorsed. The MINI-KID is the structured psychiatric interview of choice for psychiatric evaluation and outcome tracking in clinical psychopharmacology trials and epidemiological studies. In a validation study (Sheehan et al., 2010), the MINI-KID generated reliable and valid psychiatric diagnoses for children and adolescents and does so in one-third of the time as the Kiddie Schedule for Affective Disorders and Schizophrenia Present and Lifetime Version. The standard MINI-KID Version 7.0.2 for DSM-5 assesses the 30 most common and clinically relevant disorders or disorder subtypes in pediatric mental health. With this version the child and parent are interviewed together. The MINI-KID should be completed by an individual who has experience in the evaluation of pediatric patients with ADHD and the scale, and may include physicians, or licensed psychologists/clinicians. All individuals performing this assessment must be preapproved by the sponsor or designee.

#### 7.2.2 Efficacy

# 7.2.2.1 The ADHD-Rating Scale-5

The ADHD-RS-5 (DuPaul et al., 2016), the primary efficacy measure, is completed by the clinician and will be administered at baseline and each subsequent visit up to and including Visit 16/ET to capture the ADHD symptoms within each study period.

The ADHD-RS rating scale was developed to measure the behaviors of children with ADHD and is commonly used in clinical studies of ADHD (Buitelaar et al., 2007; Döpfner et al., 2006; Kratochvil et al., 2001; Michelson et al., 2001; Spencer et al., 2001). The ADHD-RS-5 consists of 18 items designed to reflect current symptomatology of ADHD based on DSM-5 criteria. Each item is scored on a 4-point scale ranging from 0 (reflecting no symptoms) to 3 (reflecting severe symptoms) with total scores ranging from 0-54. The 18 items may be grouped into 2 subscales: hyperactivity/impulsivity (9 items) and inattentiveness (9 items).

The ADHD-RS-5 should be completed by a clinician experienced in the evaluation of children with ADHD. Since the ADHD-RS-5 is an important measure for guidance in dosing decisions, the ADHD-RS-5 must be performed by an individual who is experienced with the scale. All individuals performing this assessment must be pre-approved by the sponsor or designee.

The title, version, and date of the ADHD-RS-5 used in this study are included in Table 1.

# 7.2.2.2 Clinical Global Impression

The Clinical Global Impression Scale (Guy, 1976) permits a global evaluation of the subject's severity and improvement over time.

The Clinical Global Impression has been used extensively in clinical studies of ADHD (Michelson et al., 2001; Weiss et al., 2005; Wilens et al., 2001).

For Group B, the investigator will perform the CGI-S to rate the severity of a subject's condition on a 7-point scale ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill subjects) at the baseline visit (Visit 2). Additionally at the baseline visit, the investigator should establish 3 target areas of improvement with the subject and the subject's parent/LAR. To generate the targets, an open-ended question such as "If this program of treatment works for your child, what things do you hope he/she will be doing better?" should be asked. Ratings will be completed with respect to ADHD symptoms.

For Group A and Group B, at each visit from Visit 3 up to and including Visit 16/ET, the investigator will assess the subject's improvement relative to the 3 target areas of improvement recorded at the baseline visit (Visit 2), on the CGI-I, a 7-point scale ranging from 1 (very much improved) to 7 (very much worse).

The CGI-S and CGI-I should be completed by a clinician experienced in the evaluation of children with ADHD. Since the CGI-I is an important measure for guidance in dosing decisions, the CGI-I must be performed by a principal investigator or subinvestigator who is

medically/clinically responsible for the subject and experienced with the scale. All individuals performing this assessment must be pre-approved by the sponsor or designee

The title, version, and date of the CGI-S and the CGI-I used in this study are included in Appendix 3.

# **7.2.3** Safety

The name and address of each third-party vendor (eg, clinical laboratory) used in this study will be maintained in the investigator's and sponsor's files.

# **7.2.3.1** Medical and Medication History

For subjects in Group A, any new medical history, ie, medical conditions that arose after the recording of the medical history in the antecedent study will be recorded at baseline (Visit 2).

For subjects in Group B, the investigator will take a complete medical history at the screening visit (Visit 1), including a medication history, and record all information gathered. The investigator must record all clinically or medically relevant information regardless of how much time has elapsed since the date of diagnosis.

With the consent of the subject and subject's parent/LAR, medical records from other treatment providers should be requested.

# 7.2.3.2 Physical Examination (Including Height and Weight)

For subjects in Group A, a full physical examination will be performed at the baseline visit (Visit 2) and at the end of treatment visit (Visit 16).

For subjects in Group B, a full physical examination will be performed at the screening visit (Visit 1) and at the end of treatment visit (Visit 16). Additionally, an abbreviated physical examination is required at the baseline visit (Visit 2) if >32 days have elapsed since the physical examination completed as part of the screening visit (Visit 1) was performed.

A physical examination will be performed by a qualified, licensed individual per local requirements (eg, physician, physician assistant, or nurse practitioner).

A full physical examination is composed of a review of the following body systems:

- General appearance
- Skin
- Head, eyes, ears, nose, and throat
- Spine/Neck/Thyroid
- Respiratory
- Cardiovascular
- Abdomen (including liver and kidneys)


- Musculoskeletal
- Neurological

If an abbreviated physical examination is required at the baseline visit (Visit 2), a review of the body systems will include the following:

- General appearance
- Respiratory
- Cardiovascular

For subjects in Group A, abnormalities identified at the baseline visit (Visit 2) will be documented in the subject's source documents. Changes after the baseline visit (Visit 2) will be captured as TEAEs, as determined by the investigator.

For subjects in Group B, abnormalities identified at the screening visit (Visit 1) will be documented in the subject's source documents. Changes after the screening visit (Visit 1) will be captured as TEAEs, as determined by the investigator.

#### 7.2.3.3 Adverse Event Collection

At each study visit, parent/LAR and/or subject will be questioned in a general way to ascertain if AEs have occurred since the previous visit (eg, "Have you had any health problems since your last visit?"). Adverse events are collected from the time informed consent is signed. (Refer to Section 8.) This information should be collected prior to the completion of assessments at all study visits. In addition, any symptoms/conditions reported during assessments and deemed to be clinically significant by the investigator will be assessed as AEs.

# **7.2.3.4 Vital Signs**

For subjects in Group A, measurements of oral or tympanic temperature, pulse, sitting blood pressure, and respiratory rate will be performed according to the schedule shown in Table 1. Measurement of temperature and respiratory rate will be performed as part of the last dose maintenance visit of the antecedent study.

For subjects in Group B, measurements of oral or tympanic temperature and sitting respiratory rate will be performed at the screening visit (Visit 1) only (Table 2). Measurements of sitting systolic and diastolic blood pressure and pulse will be performed at each visit to the site. Blood pressure, pulse, and respiratory rate will be determined after subjects have remained seated for a minimum of 3 minutes

Blood pressure will be determined by age-appropriate cuff (the same equipment and the same arm should be used throughout the study). A blood pressure cuff appropriate for the subject's arm length and girth should be used for all blood pressure measurements. The age-appropriate cuff should be approximately two-thirds the length/width of the subject's arm (from elbow to shoulder). All blood pressure measurements should be performed throughout the study using the age-appropriate cuff and should be performed by the same study center personnel (if possible)


throughout the study. Three measurements should be obtained using the age-appropriate cuff with at least 2 minutes in between each collection for blood pressure and pulse and report the average of the 3 measurements for each parameter. The 3 individual measurements and the averaged reading should be recorded in the source documents.

Any clinically significant deviations from baseline (Visit 2) in vital signs that are deemed clinically significant in the opinion of the investigator are to be recorded as a TEAE.

## 7.2.3.5 Height and Weight

Height will be captured at baseline and each monthly treatment visit for all subjects. A calibrated stadiometer must be used for all height measurements. Height should be measured in inches or centimeters without shoes with the subject standing on a flat surface and with chin parallel to the floor. The body should be straight but not rigid. The subject's height should be recorded as accurately as possible and should be recorded to the nearest centimeter.

Weight will be captured at each visit to the site. The same calibrated scale must be used for all weight measurements. Weight should be measured in pounds or kilograms without shoes and with light clothing. Weight should be recorded as accurately as possible and should be recorded to the nearest 0.1 pound or 0.1 kilogram.

### 7.2.3.6 Clinical Laboratory Evaluations

All clinical laboratory assays will be performed according to the laboratory's normal procedures. Reference ranges are to be supplied by the laboratory and will be used to assess the clinical laboratory data for clinical significance and out-of-range pathological changes. The investigator should assess out-of-range clinical laboratory values for clinical significance, indicating if the value(s) is/are not clinically significant or clinically significant. Abnormal clinical laboratory values, which are unexpected or not explained by the subject's clinical condition, may, at the discretion of the investigator or sponsor, be repeated as soon as possible until confirmed, explained, or resolved.

Clinical laboratory evaluations will be performed as per schedule of assessments Table 1 (Group A) and Table 2 (Group B). Additionally, for subjects in Group B, clinical laboratory tests are required to be repeated before the baseline visit (Visit 2), and the results reviewed before enrolling the subject in the study, if >32 days have elapsed since the clinical laboratory evaluations completed as part of the screening visit (Visit 1) were performed.

\*Note: Blood and urine samples may be stored for up to but not longer than 25 years.

Study Protocol Amendment 2 SHP465-308

P465-308 18 May 2018


The following clinical laboratory evaluations will be performed:

# **Biochemistry and Endocrinology**

A blood sample (~3 mL) for biochemistry will be taken to assess the following parameters:

Total cholesterol Calcium

Aspartate aminotransferase Urate

Phosphorus Blood urea nitrogen

Alanine aminotransferase Total bilirubin

Sodium Creatinine

Alkaline phosphatase Glucose

Potassium Albumin

Gamma-glutamyl transferase Total protein

Thyroid-stimulating hormone Lactate dehydrogenase

Thyroxine, Free

# Hematology

A blood sample (~2 mL) for hematology will be taken to assess the following parameters:

Hemoglobin Neutrophils

Hematocrit Lymphocytes

Red blood cells Monocytes

Platelet count Eosinophils

White blood cell count – total and differential Basophils

Mean corpuscular hemoglobin Neutrophils Band Forms

Mean corpuscular hemoglobin concentration Mean corpuscular volume

Study Protocol Amendment 2

SHP465-308 18 May 2018

# Urinalysis

A urine sample (~10 mL) for urinalysis will be collected to assess the following parameters:

Glucose pH

Specific gravity Urobilinogen

Blood Color

Ketones Leukocyte esterase

Protein Nitrite

Bilirubin

If urinalysis detects protein and/or blood, a microscopic examination will be conducted. The microscopic examination will consist of red blood cell, white blood cell, casts, and bacteria.

For Group B subjects, a urine drug and alcohol screen will be conducted at the screening visit (Visit 1). As a reminder, a urine drug screen should be repeated at the baseline visit (Visit 2) if more than 32 days have elapsed since the screening visit (Visit 1). The following drugs/drug classes will be tested:

# **Urine Drug Screen**

Cocaine Cannabinoids

Phencyclidine *d*-amphetamine

Benzodiazepines class Barbiturates class

Opiates class Propoxyphene

Methagualone Methadone

Methamphetamine

The urine drug screen must be negative at the screening visit (Visit 1) for the subject to be eligible to enroll in the study.

If the subject has a positive urine drug screen at the screening visit (Visit 1) that the investigator is able to attribute to a medication that has been prescribed to the subject, the urine drug screen must be repeated at the baseline visit (Visit 2) and must be negative so the investigator can verify that the disallowed medication which caused a positive result at the screening visit (Visit 1) has been discontinued prior to the baseline visit (Visit 2).

### 7.2.3.7 Pregnancy Test

For Group A subjects, a serum  $\beta$ -HCG pregnancy test is performed on all females of child-bearing potential at the baseline visit (Visit 2). For Group B subjects, a serum  $\beta$ -HCG

pregnancy test is performed on all females of child-bearing potential at the screening visit (Visit 1).

Additionally, the serum pregnancy test must be repeated at the baseline visit (Visit 2) if greater than 32 days have elapsed since the screening visit (Visit 1). The results must be reviewed by the investigator before the subject can be randomized.

For Group A subjects, a urine pregnancy test is performed on all females of child-bearing potential at Visit 5, and all subsequent visits until Visit 16/ET. For Group B subjects, a urine pregnancy test is performed on all females of child-bearing potential at the baseline visit (Visit 2), and all subsequent visits from Visit 5 to Visit 16/ET.

#### 7.2.3.8 Electrocardiogram

A 12-lead ECG will be performed as per schedule of assessments Table 1 (Group A) and Table 2 (Group B). Additionally, for subjects in Group B, a 12-lead ECG is required to be repeated before the baseline visit (Visit 2), and the results reviewed before enrolling the subject in the study, if >32 days have elapsed since the 12-lead ECG completed as part of the screening visit (Visit 1) was performed. Additional ECGs may be performed during the study at the investigator's discretion. Electrocardiograms will be recorded in triplicate with approximately 3 minutes apart at the screening visit or baseline visit for Group B.

All ECGs will be performed after 3 minutes of rest using the central ECG provider's equipment and will be sent to the central ECG provider electronically.

The initial interpretation of the ECG, normal or abnormal and clinical significance, will be performed immediately after collection to ensure the safety of each subject. An ECG tracing will then be evaluated by a cardiologist at a central ECG reading vendor and returned to the site with a determination of normal or abnormal. Upon review of the report from this vendor, the investigator will re-evaluate the clinical significance of the ECG while taking into consideration all other safety data available for the subject.

Although a central ECG reader is being used for this study, the eligibility of the subject is based on the investigator's assessment of the ECG. If abnormal and significant results are observed following assessment by the central reader, the investigator, in consultation with the appointed CRO medical monitor, reconfirms subject eligibility to continue.

All ECGs transmitted to the central ECG reader will be analyzed. If the central ECG reader receives multiple ECGs, the first readable ECGs will be analyzed as the scheduled ECG. Every ECG transmitted to the central ECG reader will have corresponding source document data collected. No ECG should be deleted by study site personnel. All ECGs must be transmitted to the central provider regardless of quality, results, or number of ECGs taken at a respective visit.

#### 7.2.3.9 Post Sleep Questionnaire

The PSQ is a 7-item questionnaire typically used to assess sleep quality with pharmacologic treatment. The questionnaire collects data on average time to sleep, sleep latency, frequency of interrupted sleep, duration of interrupted sleep, total sleep time and sleep quality over the last week. The PSQ will be completed by the parent/LAR with the subject and the responses will be reviewed by the clinician during the study visit.

The PSQ will be conducted at each visit to the site starting with the baseline visit (Visit 2) and will be completed by the subject's parent/LAR. The title, version, and date of the PSQ version used in this study are included in Appendix 3.

### 7.2.3.10 Children's Sleep Habits Questionnaire

The CSHQ is a tool designed to screen for the most common sleep problems in children and consists of 33 items for scoring and several extra items intended to provide administrators with other potentially useful information about respondents. The instrument evaluates the child's


sleep based on behavior within 8 different subscales: bedtime resistance, sleep-onset delay, sleep duration, sleep anxiety, night wakings, parasomnias, sleep-disordered breathing, and daytime sleepiness.

The CSHQ will be conducted at each visit to the site starting with the baseline visit (Visit 2) and will be completed by the subject's parent/LAR.

#### 7.2.3.11 Columbia-Suicide Severity Rating Scale-Baseline Version

The C-SSRS (Posner, 2007) is a semistructured interview that captures the occurrence, severity, and frequency of suicide related thoughts and behaviors during the assessment period. The interview includes definitions and suggested questions to solicit the type of information needed to determine if a suicide-related thought or behavior occurred.

The C-SSRS contains 2 required items pertaining to suicidal ideation, 4 required items pertaining to suicidal behavior, and 1 required item pertaining to nonsuicidal but self-injurious behavior. In situations where there is a positive response to the screening questions, there are 8 additional suicidal ideation items and 4 additional suicidal behavior items which are completed. Thus, there is a maximum of 19 items to be completed.

The C-SSRS must be performed by an individual who is medically responsible for the subject. All individuals performing this assessment must be preapproved by the sponsor or delegated vendor.

The Pediatric/Cognitively Impaired Version of the scale will be used in the study. Two time point versions of the C-SSRS are used in this study as follows:

- For Group B subjects only, the "baseline" version will be administered at the screening visit (Visit 1).
- For Group A and B subjects, the "since last visit" version will be completed at the baseline visit (Visit 2) and all visits afterwards.

The title, version, and date of the C-SSRS "baseline" version and the C-SSRS "since last visit" version used in this study are included in Appendix 3.

### 7.2.3.12 Suitability of the Subject to Remain in the Study

At each visit (except for Visit 16/ET) starting with the baseline visit (Visit 2), the investigator will assess the subject's ability to continue in the study. The investigator or a medically qualified designee will review all available safety information (including sleep behavior, weight and BMI) and will evaluate for the presence of insomnia or decreased appetite potentially leading to weight loss. In cases where the subject has clinically significant decreases in appetite or insomnia, the investigator should intervene as necessary based on clinical judgment (eg, diet, behavioral interventions, sleep hygiene) and consider discontinuation of treatment if necessary. In any cases where a subject has clinically significant and persistent sleep difficulties (eg, the CSHQ score of ≥41 for 2 consecutive weeks since the beginning of treatment) or has had ≥7% weight loss the investigator must discuss the case with the medical monitor and assess whether it's in the best

interest for the subject to remain in the study. The evaluation and decision should also be clearly documented in the subject's source notes.

As part of the assessment of the subject's suitability to remain in the study the investigator should also assess the subject's current potential for suicide, suicidal ideation, self-harm, or harm to others, as well as psychiatric disorders. The investigator should make this assessment by conducting a clinical interview with the subject and by reviewing of all other relevant sources available, including results of the C-SSRS. Any subject who has 1 or more positive responses must undergo further evaluation to ensure that they are not in any way at risk. As part of this assessment, if appropriate, the investigator should discuss risk factors for suicide with the subject. Where a subject has suffered an accidental injury, the investigator should ensure that this was a true accidental injury, rather than an episode of self-harming or a suicide attempt.

The investigator should pay particular attention to:

• Any 'yes' response to Items 2, 3, 4, or 5 on the C-SSRS or any suicidal behavior

The subject's source notes should clearly document that the assessment of continued suitability including assessment of the subject's appetite, weight loss, insomnia and current potential risk of suicide, suicidal ideation, feelings of hopelessness, drug use, self-harm, or harm to others has taken place and should contain the decision on whether the subject is suitable to continue in the study.

# 7.2.4 Volume of Blood to Be Drawn From Each Subject

Table 4: Volume of Blood to Be Drawn From Each Subject

| Assessment | | Sample Volume (mL) | Number of<br>Samples | Total Volume (mL) |
|---|---|---|---|---|
| Safety | Biochemistry | 3 | 3 | 9 |
| | Hematology | 2 | 3 | 6 |
| Total | | | | 15 |

During this study, it is expected that approximately 15 mL of blood will be drawn from all subjects, regardless of sex.

Note: The amount of blood to be drawn for each assessment is an estimate. The amount of blood to be drawn may vary according to the instructions provided by the manufacturer or laboratory for an individual assessment; however, the total volume drawn over the course of the study should be approximately 15 mL. When >1 blood assessment is to be done at the time point/period, if they require the same type of tube, the assessments may be combined. If a catheter is used, the first 1 mL of blood from each sampling will be discarded. For subjects in Group B, biochemistry and hematology clinical laboratory tests will be repeated at the baseline visit (Visit 2) if >32 days have elapsed since the screening visit (Visit 1).

#### 8 ADVERSE AND SERIOUS ADVERSE EVENTS ASSESSMENT

# 8.1 Definition of Adverse Events, Period of Observation, Recording of Adverse Events

An AE is any untoward medical occurrence in a clinical investigation subject administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product (ICH Guidance E2A 1995).

All AEs are collected from the time the informed consent is signed until the defined follow-up period stated in Section 7.1.3. This includes events occurring during the screening phase of the study, regardless of whether or not investigational product is administered. Where possible, a diagnosis rather than a list of symptoms should be recorded. If a diagnosis has not been made, then each symptom should be listed individually. All AEs should be captured in the source documents. In addition to untoward AEs, unexpected benefits outside the investigational product indication should also be captured.

All AEs must be followed to closure (the subject's health has returned to his/her baseline status or all variables have returned to normal), regardless of whether the subject is still participating in the study. Closure indicates that an outcome is reached, stabilization achieved (the investigator does not expect any further improvement or worsening of the event), or the event is otherwise explained. When appropriate, medical tests and examinations are performed so that resolution of event(s) can be documented.

#### 8.1.1 Severity Categorization

The severity of AEs must be recorded during the course of the event including the start and stop dates for each change in severity. An event that changes in severity should be captured as a new event. Worsening of pretreatment events, after initiation of investigational product, must be recorded as new AEs (for example, if a subject experiences mild intermittent dyspepsia before dosing of investigational product, but the dyspepsia becomes severe and more frequent after first dose of investigational product has been administered, a new AE of severe dyspepsia [with the appropriate date of onset] is recorded on the appropriate source documents).

The medical assessment of severity is determined by using the following definitions:

**Mild:** A type of AE that is usually transient and may require only minimal treatment or

therapeutic intervention. The event does not generally interfere with usual

activities of daily living.

**Moderate:** A type of AE that is usually alleviated with specific therapeutic intervention. The

event interferes with usual activities of daily living, causing discomfort but poses

no significant or permanent risk of harm to the research subject.

**Severe:** A type of AE that interrupts usual activities of daily living, or significantly affects

clinical status, or may require intensive therapeutic intervention.

# 8.1.2 Relationship Categorization

A physician/investigator must make the assessment of relationship to investigational product for each AE. The investigator should decide whether, in his or her medical judgment, there is a reasonable possibility that the event may have been caused by the investigational product. If there is no valid reason for suggesting a relationship, then the AE should be classified as "not related." Otherwise, if there is any valid reason, even if undetermined or untested, for suspecting a possible cause-and-effect relationship between the investigational product and the occurrence of the AE, then the AE should be considered "related." The causality assessment must be documented in the source documents

The following additional guidance may be helpful:

| Term | Relationship Definition |
|---|---|
| Related | The temporal relationship between the event and the administration of the investigational product is compelling and/or follows a known or suspected response pattern to that product, and the event cannot be explained by the subject's medical condition, other therapies, or accident. |
| Not Related | The event can be readily explained by other factors such as the subject's underlying medical condition, concomitant therapy, or accident and no plausible temporal or biologic relationship exists between the investigational product and the event. |

# 8.1.3 Outcome Categorization

The outcome of AEs must be recorded during the course of the study on the source documents. Outcomes are as follows:

- Fatal
- Not Recovered/Not Resolved
- Recovered/Resolved
- Recovered/Resolved With Sequelae
- Recovering/Resolving
- Unknown

# 8.1.4 Symptoms of the Disease Under Study

Symptoms of the disease under study should not be classed as AEs as long as they are within the normal day-to-day fluctuation or expected progression of the disease and are part of the efficacy data to be collected in the study; however, significant worsening of the symptoms should be recorded as an AE.

#### 8.1.5 Clinical Laboratory and Other Safety Evaluations

A change in the value of a clinical laboratory, vital sign, or ECG assessment can represent an AE if the change is clinically relevant or if, during treatment with the investigational product, a shift

of a parameter is observed from a normal value to an abnormal value, or a further worsening of an already abnormal value.

When evaluating such changes, the extent of deviation from the reference range, the duration until return to the reference range, either while continuing treatment or after the end of treatment with the investigational product, and the range of variation of the respective parameter within its reference range, must be taken into consideration.

If, at the end of the treatment phase, there are abnormal clinical laboratory, vital sign, or ECG values that were not present at the pretreatment value observed closest to the start of study treatment, further investigations should be performed until the values return to within the reference range or until a plausible explanation (eg, concomitant disease) is found for the abnormal values.

The investigator should decide, based on the above criteria and the clinical condition of a subject, whether a change in a clinical laboratory, vital sign, or ECG parameter is clinically significant and therefore represents an AE.

## 8.1.6 Pregnancy

All pregnancies are to be reported from the time informed consent is signed until the defined follow-up period stated in Section 7.1.3.

Any report of pregnancy for any female study participant or the partner of a male study participant must be reported within 24 hours to the Shire Global Drug Safety Department using the Shire Investigational and Marketed Products Pregnancy Report Form. A copy of the Shire Investigational and Marketed Products Pregnancy Report Form (and any applicable follow-up reports) must also be sent to the CRO/Shire Medical Monitor using the details specified in the emergency contact information section of the protocol. The pregnant female study participant must be withdrawn from the study.

Every effort should be made to gather information regarding the pregnancy outcome and condition of the infant. It is the responsibility of the investigator to obtain this information within 30 calendar days after the initial notification and approximately 30 calendar days post partum.

Pregnancy complications such as spontaneous abortion/miscarriage or congenital abnormality are considered SAEs and must be reported using the Shire Clinical Trial Serious Adverse Event Form. Note: An elective abortion is not considered an SAE.

In addition to the above, if the investigator determines that the pregnancy meets serious criteria, it must be reported as an SAE using the Shire Clinical Trial Serious Adverse Event Form as well as the Shire Investigational and Marketed Products Pregnancy Report Form. The test date of the first positive serum/urine  $\beta$ -HCG test or ultrasound result will determine the pregnancy onset date.

#### 8.1.7 Abuse, Misuse, Overdose, and Medication Error

Abuse, misuse, overdose, or medication error (as defined as follows) must be reported to the sponsor according to the SAE reporting procedure whether or not they result in an AE/SAE as


described in Section 8.2. Note: The 24-hour reporting requirement for SAEs does not apply to reports of abuse, misuse, overdose, or medication errors unless these result in an SAE.

The following categories are not mutually exclusive; the event can meet >1 category:

- **Abuse** Persistent or sporadic intentional intake of investigational product when used for a nonmedical purpose (eg, to alter one's state of consciousness or get high) in a manner that may be detrimental to the individual and/or society.
- **Misuse** Intentional use of investigational product other than as directed or indicated at any dose (Note: this includes a situation where the investigational product is not used as directed at the dose prescribed by the protocol).
- **Overdose** Intentional or unintentional intake of a dose of an investigational product exceeding a prespecified total daily dose of 1 capsule of the product.
- **Medication Error** An error made in prescribing, dispensing, administration, and/or use of an investigational product. For studies, medication errors are reportable to the sponsor only as defined as follows.

Cases of subjects missing doses of the investigational product are not considered reportable as medication errors.

Medication errors should be collected/reported for all products under investigation.

The administration and/or use of the unassigned treatment is/are always reportable as a medication error.

The administration and/or use of an expired investigational product should be considered as a reportable medication error.

All investigational product provided to pediatric subjects should be supervised by the parent/LAR.

#### **8.2** Serious Adverse Event Procedures

### **8.2.1** Reference Safety Information

The reference for safety information for this study is the investigator's brochure, which the sponsor has provided under separate cover to all investigators.

### **8.2.2** Reporting Procedures

All initial and follow-up SAE reports must be reported by the investigator to the Shire Global Drug Safety Department and the CRO/Shire medical monitor within 24 hours of the first awareness of the event. Note: The 24-hour reporting requirement for SAEs does not apply to reports of abuse, misuse, overdose, or medication errors (see Section 8.1.7) unless they result in an SAE.

The investigator must complete, sign, and date the Shire Clinical Study Serious Adverse Event and Nonserious AEs Required by the Protocol Form and verify the accuracy of the information recorded on the form with the corresponding source documents (Note: Source documents are not to be sent unless requested) and fax or email the form to the Shire Global Drug Safety Department.

A copy of the Shire Clinical Study Serious Adverse Event and Nonserious AEs Required by the Protocol Form (and any applicable follow-up reports) must also be sent to the CRO/Shire medical monitor using the details specified in the emergency contact information section of the protocol.

### **8.2.3** Serious Adverse Event Definition

An SAE is any untoward medical occurrence (whether considered to be related to investigational product or not) that at any dose:

- Results in death
- Is life-threatening. Note: The term "life-threatening" in the definition of "serious" refers to an event in which the subject was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it was more severe.
- Requires inpatient hospitalization or prolongation of existing hospitalization. Note: Hospitalizations, which are the result of elective or previously scheduled surgery for pre-existing conditions, which have not worsened after initiation of treatment, should not be classified as SAEs. For example, an admission for a previously scheduled ventral hernia repair would not be classified as an SAE; however, complication(s) resulting from a hospitalization for an elective or previously scheduled surgery that meet(s) serious criteria must be reported as SAE(s).
- Results in persistent or significant disability/incapacity
- Is a congenital abnormality/birth defect
- Is an important medical event. Note: Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered an SAE when, based upon appropriate medical judgment, they may jeopardize the subject and may require medical or surgical intervention to prevent 1 of the outcomes listed in this definition. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home; blood dyscrasias or convulsions that do not result in inpatient hospitalization; or the development of drug dependency or drug abuse.

#### **8.2.4** Serious Adverse Event Collection Time Frame

All SAEs (regardless of relationship to study) are collected from the time the subject signs the informed consent until the defined follow-up period stated in Section 7.1.3 and must be reported to the Shire Global Drug Safety Department and the CRO/Shire medical monitor within 24 hours of the first awareness of the event.


In addition, any SAE(s) considered "related" to the investigational product and discovered by the investigator at any interval after the study has completed must be reported to the Shire Global Drug Safety Department within 24 hours of the first awareness of the event.

#### 8.2.5 Serious Adverse Event Onset and Resolution Dates

The onset date of the SAE is defined as the date the event meets serious criteria. The resolution date is the date the event no longer meets serious criteria, the date the symptoms resolve, or the date the event is considered chronic. In the case of hospitalizations, the hospital admission and discharge dates are considered the onset and resolution dates, respectively.

In addition, any signs or symptoms experienced by the subject after signing the informed consent form, or leading up to the onset date of the SAE, or following the resolution date of the SAE, must be recorded as an AE, if appropriate.

#### **8.2.6** Fatal Outcome

Any SAE that results in the subject's death (ie, the SAE was noted as the primary cause of death) must have fatal checked as an outcome with the date of death recorded as the resolution date. For all other events ongoing at the time of death that did not contribute to the subject's death, the outcome should be considered not resolved, without a resolution date recorded.

For any SAE that results in the subject's death or any ongoing events at the time of death, unless another investigational product action was previously taken (eg, drug interrupted, reduced, withdrawn), the action taken with the investigational product should be recorded as "dose not changed" or "not applicable" (if the subject never received investigational product). The investigational product action of "withdrawn" should not be selected solely as a result of the subject's death.

# 8.2.7 Regulatory Agency, Institutional Review Board, Ethics Committee, and Site Reporting

The sponsor and clinical CRO are responsible for notifying the relevant regulatory authorities and US central IRBs of related, unexpected SAEs.

In addition the sponsor and clinical CRO are responsible for notifying active sites of all related, unexpected SAEs occurring during all interventional studies across the SHP465 program.

The investigator is responsible for notifying the local IRB, local Ethics Committee (EC), or the relevant local regulatory authority of all SAEs that occur at his or her site as required.

#### 9 DATA MANAGEMENT AND STATISTICAL METHODS

#### 9.1 Data Collection

SHP465-308

The investigators' authorized site personnel must enter the information required by the protocol on the source documents. A study monitor will visit each site in accordance with the monitoring plan and review the CRF data against the source data for completeness and accuracy. Discrepancies between source data and data entered on the CRF will be addressed by qualified site personnel. When a data discrepancy warrants correction, the correction will be made by authorized site personnel. Data collection procedures will be discussed with the site at the site initiation visit and/or at the investigator's meeting. Once a subject is randomized, it is expected that site personnel will complete the source documents entry as soon as possible to ensure data accuracy and completeness.

# 9.2 Clinical Data Management

Data are to be entered into a clinical database as specified in the CRO's data management plan. Quality control and data validation procedures are applied to ensure the validity and accuracy of the clinical database.

Data are to be reviewed and checked for omissions, errors, and values requiring further clarification using computerized and manual procedures. Data queries requiring clarification are to be communicated to the site for resolution. Only authorized personnel will make corrections to the clinical database, and all corrections are documented in an auditable manner.

# 9.3 Data Handling Considerations

Not applicable.

### 9.4 Statistical Analysis Process

The study will be analyzed by the sponsor or its agent.

The statistical analysis plan (SAP) will provide the statistical methods and definitions for the analysis of the efficacy and safety data, as well as describe the approaches to be taken for summarizing other study information such as subject disposition, demographics and baseline characteristics, investigational product exposure, and prior and concomitant medications. The SAP will also include a description of how missing, unused, and spurious data will be addressed.

To preserve the integrity of the statistical analysis and study conclusions, the SAP will be finalized before database lock.

All statistical analyses will be performed using SAS® (SAS Institute, Inc, Cary, NC 27513).

Shire Page 65 **Study Protocol Amendment 2** 

#### Planned Interim Analysis, Adaptive Design, and Data Monitoring Committee 9.5

#### 9.5.1 **Interim Analysis**

SHP465-308

After approximately 50 subjects have completed 6 months of study treatment, the database will be archived and all available safety and efficacy data will be analyzed for regulatory reporting reasons. After the 6-month data cut additional analyses will be performed, where applicable, for regulatory purposes such as subsequent safety updates and final report.

#### 9.5.2 **Data Monitoring Committee**

An external independent data monitoring committee (DMC) was set up to review the data pertaining to safety and tolerability of the study therapy for the duration of this program, which includes studies SHP465-112, SHP465-308, and SHP465-309. The DMC will review the data pertaining to safety and tolerability of the study therapy. Confidentiality of the unblinded DMC analyses is a critical concern and to address this, an unblinded independent reporting team will be identified within a CRO. The independent reporting team will have no involvement in the conduct of the study. Further details regarding the DMC can be found in the DMC charter, which will be available before the administration of investigational product.

Further details regarding the DMC can be found in the DMC charter, which will be available before the administration of investigational product.

#### 9.6 **Sample Size Calculation and Power Considerations**

Approximately 145 subjects will be enrolled into this study to ensure 60 subjects complete at least 6 months of study treatment. Subjects will enroll into this study from antecedent studies, SHP465-112 or SHP465-309 as well as de novo subjects who can be directly enrolled into this study. The sample size was established to provide long term safety data in children aged 4 to 12 years and will include at least 40 subjects aged 4-5 years at the time of informed consent in the antecedent trial or this trial, if directly enrolled.

The sample size for this study is not based on statistical considerations.

#### **Study Population** 9.7

- The screened set will include all subjects who have provided informed consent.
- The enrolled Set will consist of all subjects who have been assigned a subject identification number.
- The safety set will consist of all subjects who have taken at least 1 dose of investigational product.
- The full analysis set (FAS) will include all subjects in the safety set who completed at least 1 postdose efficacy assessment using ADHD-RS-5 total score.

#### 9.8 **Efficacy Analyses**

The FAS will be used to report the efficacy data.

The efficacy endpoint is defined as the change from baseline in the clinician-administered ADHD-RS-5 total score.

The CGI-I will be a second efficacy and used to determine the proportion of subjects with an "improved" measurement based on the CGI-S measured at baseline. The CGI-I categories of "very much improved" and "much improved" will be classified as "improved" and all other assessed categories are grouped together as "not improved."

Descriptive summary statistics will be presented by treatment group of the antecedent studies and overall for the observed efficacy variables. Observed and change from baseline in total score for the ADHD-RS-5 total score at each on-therapy treatment visit will be summarized using the number of subjects, mean, standard deviation, median, minimum, and maximum values.

The CGI-I categories of "very much improved" and "much improved" will be classified as "improved" and all other assessed categories are grouped together as "not improved."

The number and proportion of subjects with an "improved" measurement in CGI-I will be reported at each applicable postdose visit. CGI-I scores will also be summarized.

The efficacy data will be descriptively summarized for each age (4-5 years and 6-12 years), sex, race (white and non-white), and ethnicity sub-groups.

Rules for handling of missing data will be described in the SAP.

# 9.9 Safety Analyses

Safety assessments include the occurrence of TEAEs and evaluations of blood pressure, pulse, height, weight, BMI, results of clinical laboratory evaluations and ECG, sleep questionnaires (PSQ and CSHQ), and C-SSRS.

The safety set will be used to report the safety data. Safety analyses will be presented by treatment group of the antecedent studies and overall.

Adverse events will be coded using the Medical Dictionary for Regulatory Activities. Treatment emergent AEs are defined as AEs that started or deteriorated on or after the date of the first dose of investigational product, and no later than 3 days following the last dose of investigational product. The number of events, incidence, and percentage of TEAEs will be calculated overall, by system organ class, by preferred term, and by treatment group. Treatment emergent AEs will be further summarized by severity and relationship to investigational product. Adverse events related to investigational product, AEs leading to withdrawal, SAEs, and deaths will be similarly summarized/listed.

Clinical laboratory tests, vital signs, and ECG findings will be summarized by visit. Potentially clinically important findings will also be summarized or listed.

The PSQ and CSHQ will be summarized using appropriate descriptive statistics at each visit.

The C-SSRS results will be summarized and listings of the C-SSRS data will be provided for subjects with a positive response.

In addition, the safety data on TEAEs will also be descriptively summarized by treatment within each age (4-5 years and 6-12 years), sex, race (white and non-white), and ethnicity subgroup.

SHP465-308 18 May 2018

#### 10 SPONSOR'S AND INVESTIGATOR'S RESPONSIBILITIES

This study is conducted in accordance with current applicable regulations, ICH, and local ethical and legal requirements.

The name and address of each third-party vendor (eg, CRO) used in this study will be maintained in the investigator's and sponsor's files, as appropriate.

## 10.1 Sponsor's Responsibilities

## **10.1.1** Good Clinical Practice Compliance

The study sponsor and any third party to whom aspects of the study management or monitoring have been delegated will undertake their assigned roles for this study in compliance with all applicable industry regulations, ICH GCP Guideline E6 (1996) and any updates, and all applicable national and local laws and regulations.

Visits to sites are conducted by representatives of the study sponsor and/or the company organizing/managing the research on behalf of the sponsor to inspect study data, subjects' medical records, and source documents in accordance with current GCP and the respective local and (inter)national government regulations and guidelines. Records and data may additionally be reviewed by auditors or by regulatory authorities.

The sponsor ensures that local regulatory authority requirements are met before the start of the study. The sponsor (or a nominated designee) is responsible for the preparation, submission, and confirmation of receipt of any regulatory authority approvals required before release of investigational product for shipment to the site.

### **10.1.2** Public Posting of Study Information

The sponsor is responsible for posting appropriate study information on applicable websites. Information included in clinical study registries may include participating investigators' names and contact information

# 10.1.3 Submission of Summary of Clinical Study Report to Competent Authorities of Member States Concerned and Ethics Committees

The sponsor will provide a summary of the clinical study report to the competent authority of the member state(s) concerned as required by regulatory requirement(s) and to comply with the community guideline on GCP. This requirement will be fulfilled within 6 months of the end of the study completion date for pediatric studies and within 1 year for nonpediatric studies as per guidance.

## 10.1.4 Study Suspension, Termination, and Completion

The sponsor may suspend or terminate the study, or part of the study, at any time for any reason. If the study is suspended or terminated, the sponsor will ensure that applicable sites, regulatory agencies, and IRBs/ECs are notified as appropriate. Additionally, the discontinuation of a

Study Protocol Amendment 2 SHP465-308

18 May 2018


registered clinical study which has been posted to a designated public website will be updated accordingly.

#### 10.2 Investigator's Responsibilities

# 10.2.1 Good Clinical Practice Compliance

The investigator must undertake to perform the study in accordance with ICH GCP Guideline E6 (1996) and any updates, and applicable regulatory requirements and guidelines.

It is the investigator's responsibility to ensure that adequate time and appropriately trained resources are available at the site before commitment to participate in this study. The investigator should also be able to estimate or demonstrate a potential for recruiting the required number of suitable subjects within the agreed recruitment period.

The investigator will maintain a list of appropriately qualified persons to whom the investigator has delegated significant study-related tasks, and shall, upon request of the sponsor, provide documented evidence of any licenses and certifications necessary to demonstrate such qualification. Curricula vitae for investigators and subinvestigators are provided to the study sponsor (or designee) before starting the study.

If a potential research subject has a primary care physician, the investigator should, with the subject's consent, inform the physician of the subject's participation in the study.

A coordinating principal investigator is appointed to review the final clinical study report for multicenter studies. Agreement with the final clinical study report is documented by the signed and dated signature of the principal investigator (single-site study) or coordinating principal investigator (multicenter study).

# 10.2.2 Protocol Adherence and Investigator Agreement

The investigator and any coinvestigators must adhere to the protocol as detailed in this document. The investigator is responsible for enrolling only those subjects who have met protocol eligibility criteria. Investigators are required to sign an investigator agreement to confirm acceptance and willingness to comply with the study protocol.

If the investigator suspends or terminates the study at their site, the investigator will promptly inform the sponsor and the IRB/EC and provide them with a detailed written explanation. The investigator will also return all investigational product, containers, and other study materials to the sponsor. Upon study completion, the investigator will provide the sponsor, IRB/EC, and regulatory agency with final reports and summaries as required by (inter)national regulations.

Communication with local IRBs/ECs, to ensure accurate and timely information is provided at all phases during the study, may be done by the sponsor, applicable CRO, investigator, or for multicenter studies, the coordinating principal investigator according to national provisions and will be documented in the investigator agreement.

#### 10.2.3 Documentation and Retention of Records

#### **10.2.3.1** Case Report Forms

SHP465-308

Case report forms are supplied by the CRO and should be handled in accordance with instructions from the sponsor.

The investigator is responsible for maintaining adequate and accurate medical records from which accurate information is recorded onto the CRFs, which have been designed to record all observations and other data pertinent to the clinical investigation. Case report forms must be completed by the investigator or designee as stated in the site delegation log.

All data will have separate source documentation; no data will be recorded directly onto the CRF.

All data sent to the sponsor must be endorsed by the investigator.

The clinical research associate/study monitor will verify the contents against the source data per the monitoring plan. If the data are unclear or contradictory, queries are sent for corrections or verification of data.

# 10.2.3.2 Recording, Access, and Retention of Source Data and Study Documents

Original source data to be reviewed during this study will include, but are not limited to, subject's medical file, original clinical laboratory reports, and electronic diary.

All key data must be recorded in the subject's medical records.

The investigator must permit authorized representatives of the sponsor; the respective national, local, or foreign regulatory authorities; the IRB/EC; and auditors to inspect facilities and to have direct access to original source records relevant to this study, regardless of media.

The clinical research associate/study monitor (and auditors, IRB/EC, or regulatory inspectors) may check the CRF entries against the source documents. The consent form includes a statement by which the subject agrees to the monitor/auditor from the sponsor or its representatives, national or local regulatory authorities, or the IRB/EC, having access to source data (eg, subject's medical file, appointment books, original laboratory reports, X-rays).

These records must be made available within reasonable times for inspection and duplication, if required, by a properly authorized representative of any regulatory agency (eg, the US Food and Drug Administration [FDA]) or an auditor.

Essential documents must be maintained according to ICH GCP requirements and may not be destroyed without written permission from the sponsor.

# 10.2.3.3 Audit/Inspection

To ensure compliance with relevant regulations, data generated by this study must be available for inspection upon request by representatives of, for example, the US FDA (as well as other US


national and local regulatory authorities), other regulatory authorities, the sponsor or its representatives, and the IRB/EC for each site.

#### 10.2.3.4 Financial Disclosure

The investigator is required to disclose any financial arrangement during the study and for 1 year after, whereby the outcome of the study could be influenced by the value of the compensation for conducting the study, or other payments the investigator received from the sponsor. The following information is collected: any significant payments from the sponsor or subsidiaries such as a grant to fund ongoing research, compensation in the form of equipment, retainer for ongoing consultation or honoraria; any proprietary interest in investigational product; and any significant equity interest in the sponsor or subsidiaries as defined in US FDA 21 Code of Federal Regulations 54 2(b) (1998).

# 10.2.4 Compliance to all Local, State, and National Controlled-substance Biohazard and Infectious Disease Regulations and Legislation

When using controlled substances, biohazardous material, or substances for infectious diseases, the investigator must at all times comply with all local, state, and national laws pertaining to registration and reporting with the appropriate regulatory body and control and handling of such substances.

#### 10.3 Ethical Considerations

#### 10.3.1 Informed Consent

It is the responsibility of the investigator to obtain written informed consent and assent from all study subjects before any SHP465-308 study-related procedures including screening assessments. All consent and assent documentation must be in accordance with applicable regulations and GCP. Each subject or the subject's parent/LAR, as applicable, is requested to sign and date the subject informed consent form or a certified translation if applicable, after the subject has received and read (or been read) the written subject information and received an explanation of what the study involves, including but not limited to: the objectives, potential benefits and risk, inconveniences, and the subject's rights and responsibilities. A copy of the informed consent and assent documentation (ie, a complete set of subject information sheets and fully executed signature pages) must be given to the subject or the subject's parent/LAR, as applicable. This document may require translation into the local language. Signed consent forms must remain in each subject's study file and must be available for verification at any time.

Within the source documents, site personnel should document instruction of and understanding by the parent/LAR of the safe, responsible storage, and administration of investigational product to the study subject.

The principal investigator provides the sponsor with a copy of the consent form and assent form that was reviewed by the IRB/EC and received their favorable opinion/approval. A copy of the IRB/EC's written favorable opinion/approval of these documents must be provided to the sponsor before the start of the study unless it is agreed to and documented (abiding by regulatory guidelines and national provisions) before study start that another party (ie, sponsor or


coordinating principal investigator) is responsible for this action. Additionally, if the IRB/EC requires modification of the sample subject information and consent document provided by the sponsor, the documentation supporting this requirement must be provided to the sponsor.

#### 10.3.2 Institutional Review Board or Ethics Committee

It is the responsibility of the investigator to submit this protocol, the informed consent document (approved by the sponsor or their designee), relevant supporting information, and all types of subject recruitment information to the IRB/EC for review, and all must be approved before site initiation.

Responsibility for coordinating with IRBs/ECs is defined in the investigator agreement.

Prior to implementing changes in the study, the sponsor and the IRB/EC must approve any revisions of all informed consent documents and amendments to the protocol unless there is a subject safety issue.

Investigational product supplies will not be released until the CRO has received written IRB/EC approval of and copies of revised documents.

The investigator is responsible for keeping the IRB/EC appraised of the progress of the study and of any changes made to the protocol, but in any case at least once a year. For multicenter studies, this can be done by the coordinating principal investigator, according to national provisions. The investigator must also keep the local IRB/EC informed of any serious and significant AEs.

#### 10.4 Privacy and Confidentiality

All US-based sites and laboratories or entities providing support for this study, must, where applicable, comply with Health Insurance Portability and Accountability Act (HIPAA) of 1996. A site that is not a covered entity as defined by HIPAA must provide documentation of this fact to the CRO.

The confidentiality of records that may be able to identify subjects will be protected in accordance with applicable laws, regulations, and guidelines.

After subjects have consented to take part in the study, the sponsor and/or its representatives reviews their medical records and data collected during the study. These records and data may, in addition, be reviewed by others including the following: independent auditors who validate the data on behalf of the sponsor; third parties with whom the sponsor may develop, register, or market SHP465; national or local regulatory authorities; and the IRB(s)/EC(s) which gave approval for the study to proceed. The sponsor and/or its representatives accessing the records and data will take all reasonable precautions in accordance with applicable laws, regulations, and guidelines to maintain the confidentiality of subjects' identities.

Subjects are assigned a unique identifying number; however, their initials and date of birth may also be collected and used to assist the sponsor to verify the accuracy of the data (eg, to confirm that laboratory results have been assigned to the correct subject).
Ö


18 May 2018

The results of studies – containing subjects' unique identifying number, relevant medical records, and possibly initials and dates of birth – will be recorded. They may be transferred to, and used in, other countries which may not afford the same level of protection that applies within the countries where this study is conducted. The purpose of any such transfer would include: to support regulatory submissions, to conduct new data analyses to publish or present the study results, or to answer questions asked by regulatory or health authorities.

### 10.5 Study Results/Publication Policy

Shire will endeavor to publish the results of all qualifying, applicable, and covered studies according to external guidelines in a timely manner regardless of whether the outcomes are perceived as positive, neutral, or negative.

Additionally, Shire adheres to external guidelines (eg, Good Publication Practices 2) when forming a publication steering committee, which is done for large, multicenter Phase 2 through 4 and certain other studies as determined by Shire. The purpose of the publication steering committee is to act as a noncommercial body that advises or decides on dissemination of scientific study data in accordance with the scope of this policy.

All publications relating to Shire products or projects must undergo appropriate technical and intellectual property review, with Shire agreement to publish before release of information. The review is aimed at protecting the sponsor's proprietary information existing either at the commencement of the study or generated during the study. To the extent permitted by the publisher and copyright law, the principal investigator will own (or share with other authors) the copyright on his/her publications. To the extent that the principal investigator has such sole, joint or shared rights, the principal investigator grants the sponsor a perpetual, irrevocable, royalty-free license to make and distribute copies of such publications.

The term "publication" refers to any public disclosure including original research articles, review articles, oral presentations, abstracts and posters at medical congresses, journal supplements, letters to the editor, invited lectures, opinion pieces, book chapters, electronic postings on medical/scientific websites, or other disclosure of the study results, in printed, electronic, oral, or other form.

Subject to the terms of the paragraph as follows, the investigator shall have the right to publish the study results, and any background information provided by the sponsor that is necessary to include in any publication of study results, or necessary for other scholars to verify such study results. Notwithstanding the foregoing, no publication that incorporates the sponsor's confidential information shall be submitted for publication without the sponsor's prior written agreement to publish and shall be given to the sponsor for review at least 60 days before submission for publication. If requested in writing by Shire, the institution and principal investigator shall withhold submission of such publication for up to an additional 60 days to allow for filing of a patent application.

If the study is part of a multicenter study, the first publication of the study results shall be made by the sponsor in conjunction with the sponsor's presentation of a joint, multicenter publication of the compiled and analyzed study results. If such a multicenter publication is not submitted to a journal for publication by the sponsor within an 18-month period after conclusion, abandonment,

or termination of the study at all sites, or after the sponsor confirms that there shall be no multicenter study publication of the study results, an investigator may individually publish the study results from the specific site in accordance with this section. The investigator must, however, acknowledge in the publication the limitations of the single-site data being presented.

Unless otherwise required by the journal in which the publication appears, or the forum in which it is made, authorship will comply with the International Committee of Medical Journal Editors current standards. Participation as an investigator does not confer any rights to authorship of publications.


#### 11 REFERENCES

- Arnsten, A. F. 2001. Modulation of prefrontal cortical-striatal circuits: relevance to therapeutic treatments for Tourette syndrome and attention-deficit hyperactivity disorder. *Adv Neurol*, 85, 333-41.
- Bhutta, A. T. & Anand, K. J. 2002. Vulnerability of the developing brain. Neuronal mechanisms. *Clin Perinatol*, 29, 357-72.
- Brown, K. 2003. Neuroscience. New attention to ADHD genes. Science, 301, 160-1.
- Brown, T. 1996. Attention-Deficit Disorder Scales For Adolescents and Adults. The Psychological Corporation.
- Buitelaar, J. K., Michelson, D., Danckaerts, M., Gillberg, C., Spencer, T. J., Zuddas, A., Faries, D. E., Zhang, S. & Biederman, J. 2007. A randomized, double-blind study of continuation treatment for attention-deficit/hyperactivity disorder after 1 year. *Biol Psychiatry*, 61, 694-9.
- Döpfner, M., Steinhausen, H. C., Coghill, D., Dalsgaard, S., Poole, L., Ralston, S. J. & ADORE Study Group 2006. Crosscultural reliability and validity of ADHD assessed by the ADHD Rating Scale in a pan-European study. *Eur Child Adolesc Psychiatry*, 15, 146-145.
- DuPaul, G. J., Reid, R., Anastopoulos, A. D., Lambert, M., Watkins, M. & Power, T. 2016. Parent and teacher ratings of attention-deficit/hyperactivity disorder symptoms: Factor structure and normative data. *Psychol Assess*, 28, 214-25.
- Greenfield, B. & Hechman, L. 2005. Treatment of attention deficit hyperactivity disorder in adults. *Expert Rev Neurother*, 5, 107-21.
- Guy, W. (ed.) 1976. *Clinical Global Impression (CGI)*, Rockville, MD: US Department of Health, Education, and Welfare.
- Kahn, R. S., Khoury, J., Nichols, W. C. & Lanphear, B. P. 2003. Role of dopamine transporter genotype and maternal prenatal smoking in childhood hyperactive-impulsive, inattentive, and oppositional behaviors. *J Pediatr*, 143, 104-10.
- Kratochvil, C. J., Bohac, D., Harrington, M., Baker, N., May, D. & Burke, W. J. 2001. An open-label trial of tomoxetine in pediatric attention deficit hyperactivity disorder. *J Child Adolesc Psychopharmacol*, 11, 167-70.
- Kratochvil, C. J., Vaughan, B. S., Harrington, M. J. & Burke, W. J. 2003. Atomoxetine: a selective noradrenaline reuptake inhibitor for the treatment of attention-deficit/hyperactivity disorder. *Expert Opin Pharmacother*, 4, 1165-74.
- Michelson, D., Faries, D., Wernicke, J., Kelsey, D., Kendrick, K., Sallee, F. R. & Spencer, T. 2001. Atomoxetine in the treatment of children and adolescents with attention-deficit/hyperactivity disorder: a randomized, placebo-controlled, dose-response study. *Pediatrics*, 108, E83.
- NIH 2004. The fourth report on the diagnosis, evaluation, and treatment of high blood pressure in children and adolescents. *Pediatrics*, 114, 555-76.

- Ostchega, Y., Porter, K. S., Hughes, J., Dillon, C. F. & Nwankwo, T. 2011. Resting pulse rate reference data for children, adolescents, and adults: United States, 1999-2008. *Natl Health Stat Report*, 1-16.
- Posner, K. Suicidality Issues in Clinical Trials: Columbia Suicidal Adverse Event Identification in FDA Safety Analyses Division of Metabolism and Endocrinology Products Advisory Committee Meeting, Food and Drug Administration, 2007.
- Safren, S. A., Sprich, S., Chulvick, S. & Otto, M. W. 2004. Psychosocial treatments for adults with attention-deficit/hyperactivity disorder. *Psychiatr Clin North Am*, 27, 349-60.
- Sheehan, D. V., Sheehan, K. H., Shytle, R. D., Janavs, J., Bannon, Y., Rogers, J. E., Milo, K. M., Stock, S. L. & Wilkinson, B. 2010. Reliability and validity of the Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-KID). *Journal of Clinical Psychiatry*, 71, 313-26.
- Spencer, T., Biederman, J., Heiligenstein, J., Wilens, T., Faries, D., Prince, J., Faraone, S. V., Rea, J., Witcher, J. & Zervas, S. 2001. An open-label, dose-ranging study of atomoxetine in children with attention deficit hyperactivity disorder. *J Child Adolesc Psychopharmacol*, 11, 251-65.
- Wang, Y., Zheng, Y., Du, Y., Song, D. H., Shin, Y. J., Cho, S. C., Kim, B. N., Ahn, D. H., Marquez-Caraveo, M. E., Gao, H., Williams, D. W. & Levine, L. R. 2007. Atomoxetine versus methylphenidate in paediatric outpatients with attention deficit hyperactivity disorder: a randomized, double-blind comparison trial. *Aust N Z J Psychiatry*, 41, 222-30.
- Weiss, M. & Murray, C. 2003. Assessment and management of attention-deficit hyperactivity disorder in adults. *CMAJ*, 168, 715-22.
- Weiss, M., Tannock, R., Kratochvil, C., Dunn, D., Velez-Borras, J., Thomason, C., Tamura, R., Kelsey, D., Stevens, L. & Allen, A. J. 2005. A randomized, placebo-controlled study of once-daily atomoxetine in the school setting in children with ADHD. *J Am Acad Child Adolesc Psychiatry*, 44, 647-55.
- Wilens, T. E., Spencer, T. J. & Biederman, J. 2002. A review of the pharmacotherapy of adults with attention-deficit/hyperactivity disorder. *J Atten Disord*, 5, 189-202.
- Wilens, T. E., Spencer, T. J., Biederman, J., Girard, K., Doyle, R., Prince, J., Polisner, D., Solhkhah, R., Comeau, S., Monuteaux, M. C. & Parekh, A. 2001. A controlled clinical trial of bupropion for attention deficit hyperactivity disorder in adults. *Am J Psychiatry*, 158, 282-8.

## 12 APPENDICES

Study Protocol Amendment 2 SHP465-308

18 May 2018

### APPENDIX 1 PROTOCOL HISTORY

| Document | Date | Global/Country/Site Specific |
|-------------------|-------------------|------------------------------|
| Original Protocol | 11 September 2017 | Global |
| Amendment 1 | 18 May 2018 | Global |

### APPENDIX 2 DIAGNOSTIC CRITERIA/DISEASE CLASSIFICATION

#### **Appendix 2.1 DSM-5** Criteria

### A. Either (1) or (2):

(1) Six (or more) of the following symptoms of **inattention** have persisted for at least 6 months to a degree that is maladaptive and inconsistent with developmental level:

#### Inattention

- a) often fails to give close attention to details or makes careless mistakes in schoolwork, work or other activities
- b) often has difficulty sustaining attention in tasks or play activities
- c) often does not seem to listen when spoken to directly
- d) often does not follow through on instructions and fails to finish schoolwork, chores, or duties in the workplace (not due to oppositional behavior or failure to understand instructions)
- e) often has difficulty organizing tasks and activities
- f) often avoids, dislikes, or is reluctant to engage in tasks that require sustained mental effort (such as schoolwork or homework)
- g) often loses things necessary for tasks or activities (eg, toys, school assignments, pencils, books, or tools)
- h) is often easily distracted by extraneous stimuli
- i) is often forgetful in daily activities
- (2) Six (or more) of the following symptoms of **hyperactivity-impulsivity** have persisted for at least 6 months to a degree that is maladaptive and inconsistent with developmental level:

#### Hyperactivity

- (a) often fidgets with hands or feet or squirms in seat
- (b) often leaves seat in classroom or in other situations in which remaining seated is expected
- (c) often runs about or climbs excessively in situations in which it is inappropriate (in adolescents or adults, may be limited to subjective feelings of restlessness)
- (d) often has difficulty playing or engaging in leisure activities quietly
- (e) is often "on the go" or often acts as if "driven by a motor"
- (f) often talks excessively


*Impulsivity* 

- (g) often blurts out answers before questions have been completed
- (h) often has difficulty awaiting turn
- (i) often interrupts or intrudes on others (eg, butts into conversations or games)
- B. Several inattentive or hyperactive-impulsive symptoms were present prior to age 12 years.
- C. Several impairments from the symptoms are present in 2 or more settings (eg, at school [or work] and at home).
- D. There is clear evidence of clinically significant impairment in social, academic, or occupational functioning.
- E. The symptoms do not occur exclusively during the course of a Pervasive Development Disorder, Schizophrenia, or other Psychotic Disorder and are not better accounted for by another mental disorder (eg, Mood Disorder, Anxiety Disorder, Dissociative Disorder, or a Personality Disorder).

Code based on type:

### 314.01 Attention-Deficit/Hyperactivity Disorder, Combined Type:

if both Criteria A1 and A2 are met for the past 6 months

# 314.00 Attention-Deficit/Hyperactivity Disorder, Predominately Inattentive Type:

if Criterion A1 is met but Criterion A2 is not met for the past 6 months

# **314.01** Attention-Deficit/Hyperactivity Disorder, Predominately Hyperactive-Impulsive Type: if Criterion A2 is met but Criterion A1 is not met for the past 6 months

From the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition. Copyright 2013 American Psychiatric Association.

SAFER · HEALTHIER · PEOPLE

#### Boys' Stature-for-Age and Weight-for-Age Percentiles Appendix 2.2

2 to 20 years: Boys NAME \_ Stature-for-age and Weight-for-age percentiles RECORD # \_ 12 13 14 15 16 17 18 19 20 Father's Stature AGE (YEARS) Weight BMI\* Stature Date Age 190 185 Т 180 175 68-U \*To Calculate BMI: Weight (kg) + Stature (cm) + Stature (cm) x 10,000 or Weight (lb) + Stature (in) + Stature (in) x 703 170 R 66 165 in cm 64-160 160 62 62-155 155 -60 60-TAT 150 150 -58 145 -56 U 140 105-230 R -54 135 100-220 -52 95-210 130 50 200 125 48 190 120 85 180 46 80 115 170 110 75 160 42 105 70 150 40 100 65 E 140 38 95 60-130 36 90 55-120-34 50-110 -85 -32 45-100 80 -30--90 40 -80--80 35 35 -70 30 30 -60 -60 25 25 -50 50 G 20 20 40 40 15 -30 30 10 10 AGE (YEARS) lb kg kg lb 10 5 6 8 15 16 18 Published May 30, 2000 (modified 11/21/00). SOURCE: Developed by the National Center for Health Statistics in collaboration with the National Center for Chronic Disease Prevention and Health Promotion (2000). http://www.cdc.gov/growthcharts

SHP465-308

Appendix 2.3 Blood Pressure Levels for Boys by Age and Height Percentile

## Blood Pressure Levels for Boys by Age and Height Percentile

| | BP | 100 | | Systo | lic BP ( | mmHg) | | Diastolic BP (mmHg) | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Age<br>(Year) | Percentile | ← Percentile of Height → | | | | | | | | • | Perce | entile of | Height | > | |
| | 4 | 5th | 10th | 25th | 50th | 75th | 90th | 95th | 5th | 10th | 25th | 50th | 75th | 90th | 95th |
| 1 | 50th | 80 | 81 | 83 | 85 | 87 | 88 | 89 | 34 | 35 | 36 | 37 | 38 | 39 | 3 |
| | 90th | 94 | 95 | 97 | 99 | 100 | 102 | 103 | 49 | 50 | 51 | 52 | 53 | 53 | 5 |
| | 95th | 98 | 99 | 101 | 103 | 104 | 106 | 106 | 54 | 54 | 55 | 58 | 57 | 58 | 5 |
| | 99th | 105 | 106 | 108 | 110 | 112 | 113 | 114 | 61 | 62 | 63 | 64 | 65 | 66 | 6 |
| 2 | 50th | 84 | 85 | 87 | 88 | 90 | 92 | 92 | 39 | 40 | 41 | 42 | 43 | 44 | 4 |
| | 90th | 97 | 99 | 100 | 102 | 104 | 105 | 106 | 54 | 55 | 58 | 57 | 58 | 58 | 5 |
| | 95th | 101 | 102 | 104 | 106 | 108 | 109 | 110 | 59 | 59 | 60 | 61 | 62 | 63 | 6 |
| | 99th | 109 | 110 | 111 | 113 | 115 | 117 | 117 | 66 | 67 | 68 | 69 | 70 | 71 | 7 |
| 3 | 50th | 86 | 87 | 89 | 91 | 93 | 94 | 95 | 44 | 44 | 45 | 46 | 47 | 48 | 4 |
| | 90th | 100 | 101 | 103 | 105 | 107 | 108 | 109 | 59 | 59 | 60 | 61 | 62 | 63 | 6 |
| | 95th | 104 | 105 | 107 | 109 | 110 | 112 | 113 | 63 | 63 | 64 | 65 | 66 | 67 | 6 |
| | 99th | 111 | 112 | 114 | 116 | 118 | 119 | 120 | 71 | 71 | 72 | 73 | 74 | 75 | 7 |
| 4 | 50th | 88 | 89 | 91 | 93 | 95 | 96 | 97 | 47 | 48 | 49 | 50 | 51 | 51 | 5 |
| | 90th | 102 | 103 | 105 | 107 | 109 | 110 | 111 | 62 | 63 | 64 | 65 | 66 | 66 | 6 |
| | 95th | 106 | 107 | 109 | 111 | 112 | 114 | 115 | 66 | 67 | 68 | 69 | 70 | 71 | 7 |
| | 99th | 113 | 114 | 116 | 118 | 120 | 121 | 122 | 74 | 75 | 76 | 77 | 78 | 78 | 7 |
| 5 | 50th | 90 | 91 | 93 | 95 | 96 | 98 | 98 | 50 | 51 | 52 | 53 | 54 | 55 | 5 |
| | 90th | 104 | 105 | 108 | 108 | 110 | 111 | 112 | 65 | 66 | 67 | 68 | 69 | 69 | 71 |
| | 95th | 108 | 109 | 110 | 112 | 114 | 115 | 116 | 69 | 70 | 71 | 72 | 73 | 74 | 7 |
| | 99th | 115 | 116 | 118 | 120 | 121 | 123 | 123 | 77 | 78 | 79 | 80 | 81 | 81 | 8 |
| 6 | 50th | 91 | 92 | 94 | 96 | 98 | 99 | 100 | 53 | 53 | 54 | 55 | 56 | 57 | 5 |
| | 90th | 105 | 108 | 108 | 110 | 111 | 113 | 113 | 68 | 68 | 69 | 70 | 71 | 72 | 7. |
| | 95th | 109 | 110 | 112 | 114 | 115 | 117 | 117 | 72 | 72 | 73 | 74 | 75 | 76 | 7 |
| | 99th | 116 | 117 | 119 | 121 | 123 | 124 | 125 | 80 | 80 | 81 | 82 | 83 | 84 | 84 |
| 7 | 50th | 92 | 94 | 95 | 97 | 68 | 100 | 101 | 55 | 55 | 56 | 57 | 58 | 59 | 5 |
| | 90th | 106 | 107 | 109 | 111 | 113 | 114 | 115 | 70 | 70 | 71 | 72 | 73 | 74 | 7 |
| | 95th | 110 | 111 | 113 | 115 | 117 | 118 | 119 | 74 | 74 | 75 | 76 | 77 | 78 | 7 |
| | 99th | 117 | 118 | 120 | 122 | 124 | 125 | 126 | 82 | 82 | 83 | 84 | 85 | 86 | 8 |
| 8 | 50th | 94 | 95 | 97 | 99 | 100 | 102 | 102 | 56 | 57 | 58 | 59 | 60 | 60 | 6 |
| | 90th | 107 | 109 | 110 | 112 | 114 | 115 | 116 | 71 | 72 | 72 | 73 | 74 | 75 | 7 |
| | 95th | 111 | 112 | 114 | 116 | 118 | 119 | 120 | 75 | 76 | 77 | 78 | 79 | 79 | 81 |
| | 99th | 119 | 120 | 122 | 123 | 125 | 127 | 127 | 83 | 84 | 85 | 88 | 87 | 87 | 8 |
| 9 | 50th | 95 | 96 | 98 | 100 | 102 | 103 | 104 | 57 | 58 | 59 | 60 | 61 | 61 | 6: |
| | 90th | 109 | 110 | 112 | 114 | 115 | 117 | 118 | 72 | 73 | 74 | 75 | 76 | 76 | 7 |
| | 95th | 113 | 114 | 116 | 118 | 119 | 121 | 121 | 76 | 77 | 78 | 79 | 80 | 81 | 8 |
| | 99th | 120 | 121 | 123 | 125 | 127 | 128 | 129 | 84 | 85 | 86 | 87 | 88 | 88 | 81 |
| 10 | 50th | 97 | 98 | 100 | 102 | 103 | 105 | 106 | 58 | 59 | 60 | 61 | 61 | 62 | 6 |
| | 90th | 111 | 112 | 114 | 115 | 117 | 119 | 119 | 73 | 73 | 74 | 75 | 76 | 77 | 7 |
| | 95th | 115 | 116 | 117 | 119 | 121 | 122 | 123 | 77 | 78 | 79 | 80 | 81 | 81 | 83 |
| | 99th | 122 | 123 | 125 | 127 | 128 | 130 | 130 | 85 | 86 | 86 | 88 | 88 | 89 | 9 |

### Blood Pressure Levels for Boys by Age and Height Percentile (Continued)

| | BP<br>Percentile | Systolic BP (mmHg) | | | | | | | | Diastolic BP (mmHg) | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Age<br>(Year) | | SM CV | ← Percentile of Height → | | | | | | | ← Percentile of Height → | | | | | |
| | 4 | 5th | 10th | 25th | 50th | 75th | 90th | 95th | 5th | 10th | 25th | 50th | 75th | 90th | 95th |
| 11 | 50th | 99 | 100 | 102 | 104 | 105 | 107 | 107 | 59 | 59 | 60 | 61 | 62 | 63 | 63 |
| | 90th | 113 | 114 | 115 | 117 | 119 | 120 | 121 | 74 | 74 | 75 | 76 | 77 | 78 | 78 |
| | 95th | 117 | 118 | 119 | 121 | 123 | 124 | 125 | 78 | 78 | 79 | 80 | 81 | 82 | 82 |
| | 99th | 124 | 125 | 127 | 129 | 130 | 132 | 132 | 86 | 88 | 87 | 88 | 89 | 90 | 90 |
| 12 | 50th | 101 | 102 | 104 | 106 | 108 | 109 | 110 | 59 | 60 | 61 | 62 | 63 | 63 | 64 |
| | 90th | 115 | 116 | 118 | 120 | 121 | 123 | 123 | 74 | 75 | 75 | 76 | 77 | 78 | 78 |
| | 95th | 119 | 120 | 122 | 123 | 125 | 127 | 127 | 78 | 79 | 80 | 81 | 82 | 82 | 83 |
| | 99th | 126 | 127 | 129 | 131 | 133 | 134 | 135 | 86 | 87 | 88 | 89 | 90 | 90 | 91 |
| 13 | 50th | 104 | 105 | 106 | 108 | 110 | 111 | 112 | 60 | 60 | 61 | 62 | 63 | 64 | 64 |
| | 90th | 117 | 118 | 120 | 122 | 124 | 125 | 126 | 75 | 75 | 76 | 77 | 78 | 79 | 78 |
| | 95th | 121 | 122 | 124 | 126 | 128 | 129 | 130 | 79 | 79 | 80 | 81 | 82 | 83 | 83 |
| | 99th | 128 | 130 | 131 | 133 | 135 | 136 | 137 | 87 | 87 | 88 | 89 | 90 | 91 | 91 |
| 14 | 50th | 106 | 107 | 109 | 111 | 113 | 114 | 115 | 60 | 61 | 62 | 63 | 64 | 65 | 68 |
| | 90th | 120 | 121 | 123 | 125 | 126 | 128 | 128 | 75 | 76 | 77 | 78 | 79 | 79 | 80 |
| | 95th | 124 | 125 | 127 | 128 | 130 | 132 | 132 | 80 | 80 | 81 | 82 | 83 | 84 | 84 |
| | 99th | 131 | 132 | 134 | 138 | 138 | 139 | 140 | 87 | 88 | 89 | 90 | 91 | 92 | 92 |
| 15 | 50th | 109 | 110 | 112 | 113 | 115 | 117 | 117 | 61 | 62 | 63 | 64 | 65 | 66 | 66 |
| | 90th | 122 | 124 | 125 | 127 | 129 | 130 | 131 | 76 | 77 | 78 | 79 | 80 | 80 | 81 |
| | 95th | 126 | 127 | 129 | 131 | 133 | 134 | 135 | 81 | 81 | 82 | 83 | 84 | 85 | 85 |
| | 99th | 134 | 135 | 136 | 138 | 140 | 142 | 142 | 88 | 89 | 90 | 91 | 92 | 93 | 93 |
| 16 | 50th | 111 | 112 | 114 | 116 | 118 | 119 | 120 | 63 | 63 | 64 | 65 | 66 | 67 | 67 |
| | 90th | 125 | 126 | 128 | 130 | 131 | 133 | 134 | 78 | 78 | 79 | 80 | 81 | 82 | 82 |
| | 95th | 129 | 130 | 132 | 134 | 135 | 137 | 137 | 82 | 83 | 83 | 84 | 85 | 86 | 87 |
| | 99th | 136 | 137 | 139 | 141 | 143 | 144 | 145 | 90 | 90 | 91 | 92 | 93 | 94 | 94 |
| 17 | 50th | 114 | 115 | 116 | 118 | 120 | 121 | 122 | 65 | 66 | 66 | 67 | 68 | 69 | 70 |
| | 90th | 127 | 128 | 130 | 132 | 134 | 135 | 136 | 80 | 80 | 81 | 82 | 83 | 84 | 84 |
| | 95th | 131 | 132 | 134 | 138 | 138 | 139 | 140 | 84 | 85 | 86 | 87 | 87 | 88 | 89 |
| | 99th | 139 | 140 | 141 | 143 | 145 | 146 | 147 | 92 | 93 | 93 | 94 | 95 | 96 | 97 |

BP, blood pressure

For research purposes, the standard deviations in Appendix Table B–1 allow one to compute BP Z-scores and percentiles for boys with height percentiles given in Table 3 (i.e., the 5th, 10th, 26th, 50th, 75th, 90th, and 95th percentiles). These height percentiles must be converted to height Z-scores given by (5% = -1.645; 10% = -1.28; 25% = -0.68; 50% = 0; 75% = 0.68; 90% = 1.28%; 95% = 1.645) and then computed according to the methodology in steps 2–4 described in Appendix B. For children with height percentiles other than these, follow steps 1–4 as described in Appendix B.

Source: National Heart Lung and Blood Institute; May 2004 http://www.nhlbi.nih.gov/guidelines/hypertension/child\_tbl.htm

Note: To determine the eligibility of a male subject for entry in the study (based on the study inclusion criteria), first determine the percentile of height for the subject based on their age (as a whole number based on the subject's last birthday; see the Boys' Stature-for-age and Weight-for-age Percentiles). For subjects who fall between 2 height percentiles, use the lower of the 2 percentiles. Once the subject's age and height percentile for age are determined, use the table above to determine eligibility. The subject's systolic and diastolic blood pressure readings at the screening visit (Visit 1) and the baseline visit (Visit 2) must not exceed the corresponding table value (90<sup>th</sup> blood pressure percentile) for their age and height percentile.

<sup>\*</sup> The 90th percentile is 1.28 SD, 95th percentile is 1.645 SD, and the 99th percentile is 2.326 SD over the mean.

SHP465-308

#### Girls' Stature-for-Age and Weight-for-Age Percentiles Appendix 2.4

2 to 20 years: Girls NAME Stature-for-age and Weight-for-age percentiles RECORD #



Published May 30, 2000 (modified 11/21/00).

SOURCE: Developed by the National Center for Health Statistics in collaboration with the National Center for Chronic Disease Prevention and Health Promotion (2000). http://www.cdc.gov/growthcharts



SAFER · HEALTHIER · PEOPLE

**Appendix 2.5** Blood Pressure Levels for Girls by Age and Height Percentile

## Blood Pressure Levels for Girls by Age and Height Percentile

| | BP | <u> </u> | | Systo | lic BP ( | mmHg) | | Diastolic BP (mmHg) | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Age<br>(Year) | Percentile | ← Percentile of Height → | | | | | | | | ← Percentile of Height → | | | | | |
| | | 5th | 10th | 25th | 50th | 75th | 90th | 95th | 5th | 10th | 25th | 50th | 75th | 90th | 95ti |
| 1: | 50th | 83 | 84 | 85 | 86 | 88 | 89 | 90 | 38 | 39 | 39 | 40 | 41 | 41 | 4 |
| | 90th | 97 | 97 | 98 | 100 | 101 | 102 | 103 | 52 | 53 | 53 | 54 | 55 | 55 | 5 |
| | 95th | 100 | 101 | 102 | 104 | 105 | 106 | 107 | 56 | 57 | 57 | 58 | 59 | 59 | 6 |
| | 99th | 108 | 108 | 109 | 111 | 112 | 113 | 114 | 64 | 64 | 65 | 65 | 66 | 67 | 6 |
| 2 | 50th | 85 | 85 | 87 | 88 | 89 | 91 | 91 | 43 | 44 | 44 | 45 | 46 | 46 | 4 |
| | 90th | 98 | 99 | 100 | 101 | 103 | 104 | 105 | 57 | 58 | 58 | 59 | 60 | 61 | 6 |
| | 95th | 102 | 103 | 104 | 105 | 107 | 108 | 109 | 61 | 62 | 62 | 63 | 64 | 65 | 6 |
| | 99th | 109 | 110 | 111 | 112 | 114 | 115 | 116 | 69 | 69 | 70 | 70 | 71 | 72 | 7 |
| 3 | 50th | 88 | 87 | 88 | 89 | 91 | 92 | 93 | 47 | 48 | 48 | 49 | 50 | 50 | 5 |
| | 90th | 100 | 100 | 102 | 103 | 104 | 106 | 108 | 61 | 62 | 62 | 63 | 64 | 64 | 6 |
| | 95th | 104 | 104 | 105 | 107 | 108 | 109 | 110 | 65 | 86 | 66 | 67 | 88 | 68 | 6 |
| | 99th | 111 | 111 | 113 | 114 | 115 | 116 | 117 | 73 | 73 | 74 | 74 | 75 | 76 | 7 |
| 4 | 50th | 88 | 88 | 50 | 91 | 92 | 94 | 94 | 50 | 50 | -51 | 52 | 52 | 53 | - 5 |
| | 90th | 101 | 102 | 103 | 104 | 106 | 107 | 108 | 64 | 64 | 65 | 66 | 67 | 67 | 6 |
| | 95th | 105 | 106 | 107 | 108 | 110 | 111 | 112 | 68 | 68 | 69 | 70 | 71 | 71 | 7 |
| | 99th | 112 | 113 | 114 | 115 | 117 | 118 | 119 | 76 | 76 | 78 | 77 | 78 | 79 | 7 |
| 5 | 50th | 89 | 90 | 91 | 93 | 94 | 95 | 96 | 52 | 53 | 53 | 54 | 55 | 55 | 5 |
| | 90th | 103 | 103 | 105 | 106 | 107 | 109 | 109 | 66 | 67 | 67 | 68 | 69 | 69 | 7 |
| | 95th | 107 | 107 | 108 | 110 | 111 | 112 | 113 | 70 | 71 | 71 | 72 | 73 | 73 | 7 |
| | 99th | 114 | 114 | 116 | 117 | 118 | 120 | 120 | 78 | 78 | 79 | 79 | 80 | 81 | 8 |
| 6 | 50th | 91 | 92 | 93 | 94 | 96 | 97 | 98 | 54 | 54 | 55 | 56 | 56 | 57 | 5 |
| | 90th | 104 | 105 | 108 | 108 | 109 | 110 | 111 | 68 | 68 | 69 | 70 | 70 | 71 | 7 |
| | 95th | 108 | 109 | 110 | 111 | 113 | 114 | 115 | 72 | 72 | 73 | 74 | 74 | 75 | 7 |
| | 99th | 115 | 116 | 117 | 119 | 120 | 121 | 122 | 80 | 80 | 80 | 81 | 82 | 83 | 8 |
| 7 | 50th | 93 | 93 | 95 | 96 | 97 | 88 | 99 | 55 | 56 | 56 | 57 | 58 | 58 | 5 |
| | 90th | 108 | 107 | 108 | 109 | 111 | 112 | 113 | 69 | 70 | 70 | 71 | 72 | 72 | 7 |
| | 95th | 110 | 111 | 112 | 113 | 115 | 116 | 116 | 73 | 74 | 74 | 75 | 76 | 76 | 7 |
| | 99th | 117 | 118 | 119 | 120 | 122 | 123 | 124 | 81 | 81 | 82 | 82 | 83 | 84 | 8 |
| 8 | 50th | 95 | 95 | 96 | 98 | 88 | 100 | 101 | 57 | 57 | 57 | 58 | 59 | 60 | 8 |
| | 90th | 108 | 109 | 110 | 111 | 113 | 114 | 114 | 71 | 71 | 71 | 72 | 73 | 74 | 7 |
| | 95th | 112 | 112 | 114 | 115 | 116 | 118 | 118 | 75 | 75 | 75 | 76 | 77 | 78 | 7 |
| | 99th | 119 | 120 | 121 | 122 | 123 | 125 | 125 | 82 | 82 | 83 | 83 | 84 | 85 | . 8 |
| 9 | 50th | 96 | 97 | 98 | 100 | 101 | 102 | 103 | 58 | 58 | 58 | 59 | 60 | 61 | 6 |
| | 90th | 110 | 110 | 112 | 113 | 114 | 116 | 116 | 72 | 72 | 72 | 73 | 74 | 75 | 7 |
| | 95th | 114 | 114 | 115 | 117 | 118 | 119 | 120 | 76 | 76 | 76 | 77 | 78 | 79 | 7 |
| | 99th | 121 | 121 | 123 | 124 | 125 | 127 | 127 | 83 | 83 | 84 | 84 | 85 | 86 | 8 |
| 10 | 50th | 98 | 99 | 100 | 102 | 103 | 104 | 105 | 59 | 59 | 59 | 60 | 61 | 62 | 6 |
| | 90th | 112 | 112 | 114 | 115 | 116 | 118 | 118 | 73 | 73 | 73 | 74 | 75 | 76 | 7 |
| | 95th | 116 | 116 | 117 | 119 | 120 | 121 | 122 | 77 | 77 | 77 | 78 | 79 | 80 | 8 |
| | 99th | 123 | 123 | 125 | 126 | 127 | 129 | 129 | 84 | 84 | 85 | 86 | 86 | 87 | 8 |

### Blood Pressure Levels for Girls by Age and Height Percentile (Continued)

| | BP<br>Percentile | Systolic BP (mmHg) | | | | | | | | Diastolic BP (mmHg) | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Age<br>(Year) | | | ← Percentile of Height → | | | | | | | | ← Percentile of Height → | | | | |
| | | 5th | 10th | 25th | 50th | 75th | 90th | 95th | 5th | 10th | 25th | 50th | 75th | 90th | 95th |
| 11 | 50th | 100 | 101 | 102 | 103 | 105 | 106 | 107 | 60 | 60 | 60 | 61 | 62 | 63 | 63 |
| | 90th | 114 | 114 | 116 | 117 | 118 | 119 | 120 | 74 | 74 | 74 | 75 | 76 | 77 | 77 |
| | 95th | 118 | 118 | 119 | 121 | 122 | 123 | 124 | 78 | 78 | 78 | 79 | 80 | 81 | 81 |
| | 99th | 125 | 125 | 126 | 128 | 129 | 130 | 131 | 85 | 85 | 86 | 87 | 87 | 88 | 88 |
| 12 | 50th | 102 | 103 | 104 | 105 | 107 | 108 | 109 | 61 | 61 | 61 | 62 | 63 | 64 | 64 |
| | 90th | 116 | 116 | 117 | 119 | 120 | 121 | 122 | 75 | 75 | 75 | 76 | 77 | 78 | 78 |
| | 95th | 119 | 120 | 121 | 123 | 124 | 125 | 126 | 79 | 79 | 79 | 80 | 81 | 82 | 82 |
| | 99th | 127 | 127 | 128 | 130 | 131 | 132 | 133 | 86 | 86 | 87 | 88 | 88 | 89 | 90 |
| 13 | 50th | 104 | 105 | 106 | 107 | 109 | 110 | 110 | 62 | 62 | 62 | 63 | 64 | 65 | 65 |
| | 90th | 117 | 118 | 119 | 121 | 122 | 123 | 124 | 76 | 78 | 76 | 77 | 78 | 79 | 78 |
| | 95th | 121 | 122 | 123 | 124 | 126 | 127 | 128 | 80 | 80 | 80 | 81 | 82 | 83 | 83 |
| | 99th | 128 | 129 | 130 | 132 | 133 | 134 | 135 | 87 | 87 | 88 | 89 | 89 | 90 | 9 |
| 14 | 50th | 106 | 106 | 107 | 109 | 110 | 111 | 112 | 63 | 63 | 63 | 64 | 65 | 66 | 66 |
| | 90th | 119 | 120 | 121 | 122 | 124 | 125 | 125 | 77 | 77 | 77 | 78 | 79 | 80 | 80 |
| | 95th | 123 | 123 | 125 | 126 | 127 | 129 | 129 | 81 | 81 | 81 | 82 | 83 | 84 | 84 |
| | 99th | 130 | 131 | 132 | 133 | 135 | 136 | 138 | 88 | 88 | 89 | 90 | 90 | 91 | 93 |
| 15 | 50th | 107 | 108 | 109 | 110 | 111 | 113 | 113 | 64 | 64 | 64 | 65 | 66 | 67 | 6 |
| | 90th | 120 | 121 | 122 | 123 | 125 | 126 | 127 | 78 | 78 | 78 | 79 | 80 | 81 | 8 |
| | 95th | 124 | 125 | 126 | 127 | 129 | 130 | 131 | 82 | 82 | 82 | 83 | 84 | 85 | 88 |
| | 99th | 131 | 132 | 133 | 134 | 136 | 137 | 138 | 89 | 89 | 90 | 91 | 91 | 92 | 93 |
| 16 | 50th | 108 | 108 | 110 | 111 | 112 | 114 | 114 | 64 | 64 | 65 | 66 | 66 | 67 | 68 |
| | 90th | 121 | 122 | 123 | 124 | 126 | 127 | 128 | 78 | 78 | 79 | 80 | 81 | 81 | 83 |
| | 95th | 125 | 126 | 127 | 128 | 130 | 131 | 132 | 82 | 82 | 83 | 84 | 85 | 85 | 86 |
| | 99th | 132 | 133 | 134 | 135 | 137 | 138 | 139 | 90 | 90 | 90 | 91 | 92 | 93 | 93 |
| 17 | 50th | 108 | 109 | 110 | 111 | 113 | 114 | 115 | 64 | 65 | 65 | 66 | 67 | 67 | 68 |
| | 90th | 122 | 122 | 123 | 125 | 126 | 127 | 128 | 78 | 79 | 79 | 80 | 81 | 81 | 8: |
| | 95th | 125 | 126 | 127 | 129 | 130 | 131 | 132 | 82 | 83 | 83 | 84 | 85 | 85 | 86 |
| | 99th | 133 | 133 | 134 | 136 | 137 | 138 | 139 | 90 | 90 | 91 | 91 | 92 | 93 | 93 |

BP, blood pressure

For research purposes, the standard deviations in Appendix Table B–1 allow one to compute BP Z-scores and percentiles for girls with height percentiles given in Table 4 (i.e., the 5th, 10th, 25th, 50th, 75th, 90th, and 95th percentiles). These height percentiles must be converted to height Z-scores given by (5% = -1.645; 10% = -1.28; 25% = -0.68; 50% = 0; 75% = 0.68; 90% = 1.28%; 95% = 1.645) and then computed according to the methodology in steps 2–4 described in Appendix B. For children with height percentiles other than these, follow steps 1–4 as described in Appendix B.

Source: National Heart Lung and Blood Institute; May 2004 http://www.nhlbi.nih.gov/guidelines/hypertension/child\_tbl.htm

Note: To determine the eligibility of a female subject for entry in the study (based on study inclusion criteria), first determine the percentile of height for the subject based on their age (as a whole number based on the subject's last birthday; see the Girls' Stature-for-age and Weight Percentiles). For subjects who fall between 2 height percentiles, use the lower of the 2 percentiles. Once the subject's age and height percentile for age are determined, use the table above to determine eligibility. The subject's systolic and diastolic blood pressure readings at the screening visit (Visit 1) and the baseline visit (Visit 2) must not exceed the corresponding table value (90<sup>th</sup> blood pressure percentile) for their age and height percentile.

<sup>\*</sup> The 90th percentile is 1.28 SD, 95th percentile is 1.645 SD, and the 99th percentile is 2.326 SD over the mean.

### APPENDIX 3 SCALES AND ASSESSMENTS

The following scales/assessments will be utilized in this study:

| Full Title of Scale/Assessment | Version Number | Date Issued |
|---|---|---|
| ADHD-RS-5 Child, Home Version | N/A | 2016 |
| CGI-I and CGI-S | N/A | 1976 |
| C-SSRS | Baseline | Baseline 23 Jun 2010 |
| | Since Last Visit | Since Last Visit 23 Jun 2010 |
| CSHQ | N/A | 2009 |
| MINI-KID | 7.0.2 | 08 Aug 2016 |
| PSQ | N/A | N/A |

ADHD-RS-5= Attention-deficit/Hyperactivity Disorder Rating Scale 5; CGI-I= Clinical Global Impressions – Improvement; CGI-S= Clinical Global Impressions – Severity of Illness; CSHQ=Children's Sleep Habits Questionnaire; C-SSRS= Columbia-Suicide Severity Rating Scale MINI-KID=Mini International Neuropsychiatric Interview for Children and Adolescents; N/A=not applicable; PSQ=Post Sleep Questionnaire.

A separate master file containing each scale/assessment listed above will be provided to the site. Updates to scales/assessments during the study (if applicable) will be documented in the table above and a new master file containing the revised scale/assessment will be provided to the site.